



# STATISTICAL ANALYSIS PLAN

Study CRO-PK-22-363 - Sponsor code PNET-22-08

A phase I, open label, single dose, two parts study in male and female healthy subjects to assess the safety and pharmacokinetics of Fosnetupitant 235 mg administered as IV bolus and of derived Netupitant and Netupitant metabolites

Sponsor: Helsinn Healthcare SA - Via Pian Scairolo 9,

CH-6912 Lugano - Switzerland

Phone: +41 91 985 21 21 Fax: +41 91 993 21 22

NCT number: NCT06840769

Document date: 18JUN2024



# STATISTICAL ANALYSIS PLAN

Study CRO-PK-22-363 - Sponsor code PNET-22-08

A phase I, open label, single dose, two parts study in male and female healthy subjects to assess the safety and pharmacokinetics of Fosnetupitant 235 mg administered as IV bolus and of derived Netupitant and Netupitant metabolites

Open label, single dose, two parts (part A and part B), safety and pharmacokinetics phase I study. Study Part B will be conducted according to a randomized cross-over design

Investigational product: IV fosnetupitant 235 mg free base 20 mL ready to use solution for

intravenous administration, Patheon Italia S.p.A., Italy

Reference product: IV Akynzeo (235 mg fosnetupitant/0.25 mg palonosetron) in 20 mL

injectable solution, Baxter Oncology GmbH, Germany

Placebo: 0.9% sodium chloride injection solution ready to use solution for

intravenous administration (placebo), purchased from the market

Sponsor: Helsinn Healthcare SA - Via Pian Scairolo 9,

CH-6912 Lugano - Switzerland

Phone: +41 91 985 21 21 Fax: +41 91 993 21 22

Investigator: Milko Radicioni, MD - Principal Investigator

CROSS Research S.A., Phase I Unit, Via F. A. Giorgioli 14

CH-6864 Arzo, Switzerland Phone: +41.91.64.04.450 Fax: +41.91.64.04.451

Email: clinic@croalliance.com

Development phase: Phase I

Version and date: Final version 1.0, 18JUN2024

This study will be conducted in compliance with the protocol and the principles of Good Clinical Practice (GCP) [ICH topic E6 (R2)] and with the local regulatory requirements

Property of the sponsor

May not be used, divulged, published or otherwise disclosed without the consent of the sponsor

This document comprises 31 pages plus appendices



# **VERSIONS' HISTORY**

| Version | Date of Issue | Reason for change |
|---|---|---|
| Draft version 0.1 | 22NOV2023 | issued the first draft |
| Draft version 0.2 | 10JUN2024 | issued the draft version 0.2 after Sponsor's revision |
| Final version 1.0 | 18JUN2024 | issued the final version after MW's revision |



**SPONSOR** 

Statistical analysis plan CRO-PK-22-363 Sponsor code PNET-22-08 Netupitant IV infusion shortening Final version 1.0, 18JUN2024

# APPROVAL AND ACKNOWLEDGEMENT

| Helsinn Healthcare SA |
|------------------------------------------------|
| Head of Clinical Affairs, Technical Operations |
| Head of Data Science, Technical Operations |



| CRO | | | |
|--------------|----------|-------|-------------|
| <b>CROSS</b> | Research | S.A., | Switzerland |

| Biometry Unit Representative (for approval and acknowledgement) |
|-----------------------------------------------------------------------|
| Medical Writer Team Representative (for approval and acknowledgement) |
| Coordination (for acknowledgement only) |

CROSS Research S.A.

Page 4



#### STUDY SCHEDULE

#### Study procedures of Part A

| ACTIVITIES | Screening | Admission | Active treatment administration | Observation and release | Final visit or ETV <sup>8</sup> |
|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | | V4 or ETV <sup>8</sup> |
| Day | -21 to -2 | -1 | 1 | 2 | 7 |
| Informed consent | X | | | | |
| Inclusion/Exclusion<br>criteria | X | X | | | |
| Full physical examination | X | | | | X |
| Short physical examination | | x <sup>1</sup> | | X | |
| Demographics | X | | | | |
| Medical and surgical history | X | | | | |
| Previous and concomitant treatments | x | X | X | X | x |
| Height and body mass index (BMI) | X | | | | |
| Body weight | X | X | | | X |
| Safety laboratory<br>(hematology, blood | X | | | | X |
| chemistry, urinalysis) Virology (HBs Ag, HCV Ab, HIV) | X | | | | |
| Pregnancy test | x <sup>2</sup> | x <sup>3</sup> | | | x <sup>3</sup> |
| Urine drug screen | X | X | | | |
| Salivary alcohol test | | X | | | |
| Triplicate 12-lead ECGs | X | | x <sup>4</sup> | x <sup>6</sup> | X |
| Vital signs | X | X | x <sup>5</sup> | x <sup>6</sup> | X |
| Enrolment | | X | | | |
| Confinement | | X | X | | |
| Active Treatment administration | | | x | | |
| PK blood sampling <sup>7</sup> | | | x x | | |
| Discharge | | | | X | |
| AE recording <sup>9</sup> | X | X | X | X | X |

- 1. Only if screening full physical examination performed more than 7 days before Day -1
- 2. Women only serum b-HCG test
- 3. Women only urine test
- 4. At pre-dose, at the end of injection, then at 1, 2, 4 and 24 h after end of administration; to be measured after 5 min at rest in supine position before recording.
- 5. At pre-dose, at the end of the injection, then at 1, 2, 4 and 24 h after the end of the injection; to be measured after 5 min at rest in sitting position before measurement.
- 6. Upon discharge at 24 h after the end of active treatment injection.
- 7. See schedule in tabular format at next page.
- 8. Early termination visit (ETV) upon discontinuation in case of premature termination
- 9. AEs monitored starting at the screening visit, immediately after informed consent, up to the final visit or ETV



# Schedule of PK blood sampling

| | | | Blood | sampling | g times af | ter the st | art of T | or R treat | ment | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | T injection of | | | | | | | Reference product infusion of | |
| | 2 n | nin | 5 n | nin | 15 min | | 30 min | | 30 min | 30 min |
| | Part | Part | Part | Part | Part | Part | Part | Part | Part | Part |
| | A | В | A | В | A | В | A | В | A (Rα) | B (R) |
| Pre-dose | X | X | X | X | X | X | X | X | X | X |
| 2 min | X | X | | | | | | | | |
| 5 min | X | X | X | X | | | | | | |
| 10 min | X | X | X | X | | | | | | |
| 15 min | X | X | X | X | X | X | | | | |
| 20 min | X | X | X | X | X | X | | | | |
| 30 min | X | X | X | X | X | X | X | X | X | X |
| 45 min | X | X | X | X | X | X | X | X | X | X |
| 1 h | X | X | X | X | X | X | X | X | X | X |
| 1.5 h | X | X | X | X | X | X | X | X | X | X |
| 2 h | X | X | X | X | X | X | X | X | X | X |
| 3 h | X | X | X | X | X | X | X | X | X | X |
| 4 h | X | X | X | X | X | X | X | X | X | X |
| 8 h | X | X | X | X | X | X | X | X | X | X |
| 12 h | X | X | X | X | X | X | X | X | X | X |
| 24 h | X | X | X | X | X | X | X | X | X | X |
| 48 h | | X | | X | | X | | X | | X |
| 72 h | | X | | X | | X | | X | | X |
| 96 h | | X | | X | | X | | X | | X |
| 120 h | | X | | X | | X | | X | | X |
| 144 h | | X | | X | | X | | X | | X |
| 168 h | | X | | X | | X | | X | | X |
| 192 h | | X | | X | | X | | X | | X |
| 216 h | | X | | X | | X | | X | | X |
| 240 h | | X | | X | | X | | X | | X |



# TABLES OF CONTENTS

| | STATISTICAL ANALYSIS PLAN | 1 |
|---|---|---|
| | VERSIONS' HISTORY | 2 |
| | APPROVAL AND ACKNOWLEDGEMENT | 3 |
| | STUDY SCHEDULE | 5 |
| | TABLES OF CONTENTS | 7 |
| | ABBREVIATIONS | 9 |
| 1 | INTRODUCTION | 11 |
| 1.1 | Changes with respect to the study protocol | 11 |
| 2 | STUDY OBJECTIVES | 12 |
| 2.1 | Primary end-points | 12 |
| 2.2 | Secondary safety end-points | 12 |
| 2.3 | Secondary PK end-points | 12 |
| 3 | INVESTIGATIONAL PLAN | 13 |
| 3.1 | Overall study design | 13 |
| 3.2 | Discussion of design | 13 |
| 4 | STUDY POPULATION | 14 |
| 4.1 | Target population | 14 |
| 4.2 | Inclusion criteria | 14 |
| 4.3 | Exclusion criteria | 15 |
| 4.3.1 | Not allowed treatments | 16 |
| 4.4 | Use of contraceptive methods | 16 |
| 5 | STUDY SCHEDULE | 17 |
| 5.1 | Study visits and procedures | 17 |
| 5.2 | Decisional process for escalation to next administration duration | 20 |
| 5.2.1 | Decisional process for treatment of subjects within the cohorts | 20 |
| 5.2.2 | Decisional process for escalation to next administration duration | 20 |
| 5.3 | Diet and lifestyle | 21 |
| 5.4 | Restrictions | 21 |
| 6 | STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD | 22 |
| 6.1 | Unique subject identifier | 22 |
| 6.2 | Subject identifier for the study | 22 |
| 6.3 | Randomisation | 22 |
| 6.4 | Treatment allocation | 22 |
| 6.5 | Blinding | 22 |
| 7 | STUDY EVALUATION PARAMETERS | 23 |
| 7.1 | Study variables | 23 |
| 7.1.1 | Primary safety variables | 23 |
| 7.1.2 | Secondary safety variables | 23 |
| 7.2 | PK parameters | 23 |
| 8 | STATISTICAL METHOD | 24 |
| 8.1 | Tables, listings and figures layout | 24 |
| 8.2 | Analysis sets | 25 |
| 8.2.1 | Definitions | 25 |
| 8.2.2 | Reasons for exclusion from the PK Set | 25 |




Statistical analysis plan CRO-PK-22-363 Sponsor code PNET-22-08 Netupitant IV infusion shortening Final version 1.0, 18JUN2024

| 8.3 | Sample size and power considerations | 25 |
|------------|-----------------------------------------------------------|----|
| 8.4 | Demographic, baseline and background characteristics | 26 |
| 8.4.1 | Subjects' disposition | 26 |
| 8.4.2 | <b>Analysis sets</b> | 26 |
| 8.4.3 | Subjects excluded from PK and/or safety analysis | 26 |
| 8.4.4 | Discontinued subjects | 26 |
| 8.4.5 | Protocol deviations | 26 |
| 8.4.6 | Demography | 26 |
| 8.4.7 | Physical examination | 26 |
| 8.4.8 | Fertility status and contraceptive method | 27 |
| 8.4.9 | Reproductive status and contraception | 27 |
| 8.4.10 | Salivary alcohol test, pregnancy test and urine drug test | 27 |
| 8.4.11 | Inclusion/exclusion criteria not met | 27 |
| 8.4.12 | Medical and surgical history | 27 |
| 8.4.13 | Prior and concomitant medication | 27 |
| 8.4.14 | Tobacco, alcohol and caffeine consumption | 27 |
| 8.4.15 | Subjects' study visits | 27 |
| 8.4.16 | Meals | 27 |
| 8.5 | IMP administration | 27 |
| 8.5.1 | IMP administration (date/time) | 27 |
| 8.5.2 | Fasting condition | 28 |
| 8.5.3 | Dose per body weight | 28 |
| 8.6 | PK analysis | 28 |
| 8.6.1 | PK blood samples collection | 28 |
| 8.6.2 | Descriptive pharmacokinetics | 28 |
| <b>8.7</b> | Safety and tolerability analysis | 28 |
| 8.7.1 | Adverse events | 28 |
| 8.7.2 | Vital signs | 29 |
| 8.7.3 | Body weight | 29 |
| 8.7.4 | ECG | 29 |
| 8.7.5 | Laboratory data | 30 |
| 8.7.6 | Physical examination | 30 |
| 8.8 | Analysis datasets | 30 |
| 9 | REFERENCES | 31 |
| 10 | APPENDICES | 32 |



#### **ABBREVIATIONS**

β-HCG human chorionic gonadotropin β

AE Adverse Event

AUC $_{0-t}$  Area under the concentration-time curve from time zero to time t AUC $\infty$  Area under the concentration versus time curve up to infinity

%AUCextra Percentage of the residual area extrapolated to infinity in relation to the AUC∞

BLQL Below Lower Quantification Limit

BP Blood Pressure

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval
C<sub>max</sub> Peak drug concentration
CPL Clinical Project Leader
CRF Case Report Form

CRO Contract Research Organisation

CV Coefficient of Variation
DIABP Diastolic Blood Pressure
ECG Electrocardiogram
ETV Early Termination Visit
FSFV First Subject First Visit
GCP Good Clinical Practice
GLP Good Laboratory Practice

HBs Ag Hepatitis B virus surface antigen HCV Ab Hepatitis C virus antibodies HIV Human Immunodeficiency Virus

HR Heart Rate

ICH International Conference on Harmonisation

IGA Investigator Global Assessment
IMP Investigational Medicinal Product

LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

N Normal

NA Not Applicable NC Not calculated

NCS Not clinically significant

NSAIDs Non-Steroidal Anti-Inflammatory Drugs

OTC Over The Counter
PD Pharmacodynamics
PK Pharmacokinetics
PT Preferred Term

PTAE Pre-Treatment Adverse Event

QOL Quality of Life

SYSBP Systolic Blood Pressure SD Standard Deviation SOC System Organ Class

SDTM Study Data Tabulation Model

T Test

TEAE Treatment-Emergent Adverse Event

t<sub>1/2</sub> Half-life




Statistical analysis plan CRO-PK-22-363 Sponsor code PNET-22-08 Netupitant IV infusion shortening Final version 1.0, 18JUN2024

T<sub>max</sub> Time to achieve Cmax

USDA United States Department of Agriculture

WHODDE World Health Organisation Drug Dictionary Enhanced



#### 1 INTRODUCTION

Statistical analysis is performed by the CROSS Research Biometry Unit. The end-points and methods of analysis specified in this SAP are consistent with ICH E6 (R2) and E9 guidelines (1, 2). The present SAP has been compiled for part A of the study by the CRO Biometry Unit based on the final version 3.0 of the clinical study protocol (3), reviewed by the Sponsor and finalized before the database lock.

## 1.1 Changes with respect to the study protocol

No change with respect to the study protocol (3) was introduced in this SAP.



#### 2 STUDY OBJECTIVES

The primary objective is to define the shortest safe and tolerable duration of IV injection of fosnetupitant 235 mg among 4 durations tested in decreasing order: 30, 15, 5 and 2 min, respectively.

The secondary objectives are:

- to characterize the pharmacokinetic (PK) profile in plasma of fosnetupitant, netupitant and netupitant metabolites M1, M2 and M3 after injection of T administered at the relevant injection duration and after injection of undiluted R (defined as Rα)
- to determine the safety and tolerability of T administered at the relevant injection duration

# 2.1 Primary end-points

• Type, number and frequency of TEAEs collected up to 24 h post-dose.

# 2.2 Secondary safety end-points

• Vital signs (blood pressure, pulse rate), 12-lead ECG, clinical laboratory tests (blood chemistry, hematology and urinalysis), body weight and physical examination

## 2.3 Secondary PK end-points

For plasma fosnetupitant, netupitant and its main metabolites M1, M2 and M3, when applicable the following parameters will be measured/calculated:

• C0, Cmax, tmax, Clast, tlast, AUC0-t (for all analytes), AUC0-24, λz, t½, CL, Vz, MRT



#### 3 INVESTIGATIONAL PLAN

# 3.1 Overall study design

Open label, single dose, safety and PK phase I study.

## 3.2 Discussion of design

The study design is in compliance with the relevant FDA guidance document for industry on bioavailability studies (4).

The study design is based upon that of a previous study of CINVANTI® (aprepitant injectable emulsion) published by Ottoboni et al. (5) where it is described that, due to a shortage of small volume parental solutions, the American Society of Health-System Pharmacists recommended switching the delivery of treatments from infusion to IV push.

The selected dose for the fosnetupitant component is 235 mg, corresponding to 260 mg of fosnetupitant chloride hydrochloride, previously shown to be equivalent in exposure (Netupitant AUC) to the netupitant dose present in the oral NEPA FDC (300 mg of netupitant).

See paragraph 11.2 of the study protocol (3) for further details.



#### 4 STUDY POPULATION

# 4.1 Target population

Male and female adult healthy volunteers aged between 18 and 55 years old.

#### 4.2 Inclusion criteria

To be enrolled in this study, subjects must fulfil all these criteria:

- 1. Informed consent: signed written informed consent before inclusion in the study
- 2. Sex and Age: healthy men/women volunteers, 18-55 years old (inclusive)
- 3. Body Mass Index (BMI): 18.5-30 kg/m<sup>2</sup> inclusive
- 4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, pulse rate 50-99 bpm, measured after 5 min at rest in the sitting position
- 5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
- 6. Contraception and fertility (women only): women of childbearing potential defined as a non-menopausal woman who has not had a bilateral oophorectomy or medically documented ovarian failure and/or at risk for pregnancy must agree, signing the informed consent form, to use a highly effective method of contraception throughout the study and to continue for 14 days after the last dose of the study treatment. Highly effective contraceptive measures include:
  - a. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit.
  - b. A non-hormonal intrauterine device [IUD] for at least 2 months before the screening visit
  - c. A sterile or vasectomized sexual partner
  - d. True (long-term) heterosexual abstinence, defined as refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject, while periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), lactational amenorrhea and withdrawal are not acceptable.

Women of non-child-bearing potential or in post-menopausal status defined as such when there is either:

- a. 12 months of spontaneous amenorrhea or
- b. 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or
- c. 6 weeks documented postsurgical bilateral oophorectomy with or without hysterectomy

will be admitted.

For all women, pregnancy test result must be negative at screening and admission (Day - 1).



- 7. Contraception (men only): men will either be sterile or agree to use one of the following approved methods of contraception from the first study drug administration until at least 14 days after the last administration, also in case their partner is currently pregnant:
  - a. A male condom with spermicide
  - b. A sterile sexual partner or a partner in post-menopausal status for at least one year
  - c. Use by the female sexual partner of an IUD, a female condom with spermicide, a contraceptive sponge with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, or hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit

Men must accept to inform their partners of the participation in the clinical study. Furthermore, they will not donate sperm from the date of the informed consent form's signature, throughout the study, and for at least 14 days after the last dose of the study treatment. These requirements are based upon the availability and results of reproductive toxicity data.

#### 4.3 Exclusion criteria

Subjects meeting any of these criteria will not be enrolled in the study:

- 1. 12-leads Electrocardiogram (ECG) (supine position): clinically significant abnormalities at screening. With regards to QTc, the following will be considered as exclusion criterion: mean corrected QT (QTcF) > 450 ms. HR < 50 or > 99 bpm. PR < 100 or >220 ms. QRS > 120 ms. Relevantly abnormal T-wave patterns
- 2. Physical examination findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
- 3. Laboratory analyses: clinically significant abnormal laboratory values at screening, indicative of physical illness or suggesting the subject's exclusion, in his/her best interest
- 4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
- 5. Diseases: significant history, in the opinion of the Investigator, of renal, hepatic, gastrointestinal, cardiovascular (in particular, heart failure, hypokalemia, family history of Long QT Syndrome, history of superficial thrombophlebitis or deep vein thrombosis), respiratory, skin, hematological, endocrine or neurological diseases that may interfere with the aim of the study
- 6. *Medications*: medications, including over the counter (OTC) medications and herbal remedies in the 2 weeks before the first visit of the study. Hormonal contraceptives for women are allowed
- 7. CYP3A4 inducers and inhibitors: use of any inducer or inhibitor of CYP3A4 enzymes (drugs, food, herbal remedies) in the 28 days or in the 7 days, respectively, before the planned first study drug administration and during the whole study
- 8. *Investigative drug studies*: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study



- 9. Blood donation or significant blood loss: blood donations or significant blood loss in the 3 months before the first visit of this study
- 10. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for women and >2 drinks/day for men, defined according to the USDA Dietary Guidelines 2020-2025 (317)], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
- 11. Drug test: positive result at the urine drug screening test at screening or Day -1
- 12. Alcohol test: positive salivary alcohol test at Day -1
- 13. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before screening; vegetarians
- 14. Pregnancy (women only): positive or missing pregnancy test at screening or Day -1, pregnant or lactating women
- 15. Netupitant studies: enrolment in a previous study of netupitant or fosnetupitant (alone or in combination with palonosetron)

#### 4.3.1 Not allowed treatments

No medication, including OTC and herbal remedies, will be allowed in the 2 weeks before the first visit of the study (Screening - Visit 1) and during the whole study duration. In particular, the use of CYP3A4 inducers or CYP3A4 inhibitors (drugs, food, herbs) in the 28 days or in the 7 days, respectively, before the 1<sup>st</sup> study treatment intake on Day 1 will not be allowed.

Paracetamol will be allowed as therapeutic countermeasure for certain types of AEs according to the Investigator's opinion. Hormonal contraceptives will be allowed.

The intake of any other medication will be reported as a protocol deviation. However, it will lead to subject's discontinuation from the study only if the Investigator, together with the Sponsor, considers the medication as being able to affect the study assessments or outcome.

#### 4.4 Use of contraceptive methods

In case of men or women of childbearing potential, the Investigator, in consultation with the subject, will select the appropriate method/methods of contraception for the individual according to the list of contraception methods of inclusion criteria 6 and 7, and instruct the subject or a screened man referring to his partner in their consistent and correct use. Highly effective contraceptive measures include those listed in inclusion criteria 6 and 7.

Moreover, men will not donate sperm from the date of the informed consent form's signature, throughout the study, and for at least 14 days after the last dose of the study treatment.

At screening and at each study visit, the Investigator will instruct subjects on the need to use contraception throughout the study and to continue for 14 days after the last dose of assigned treatment. In addition, the Investigator will instruct the subjects to call immediately if a selected birth control method is discontinued or if pregnancy is known or suspected.



#### 5 STUDY SCHEDULE

The schedule of the study is summarised at page 6.

#### 5.1 Study visits and procedures

Each subject will undergo 4 visits.

Study foresees, after the screening process, a confinement of approximately one and a half days at the Phase I Unit and one ambulatory visit (V4) 7 days post-dose. The maximum study duration for study will be 28 days, including the screening period.

The first subject first visit (FSFV) is defined as the 1st screening visit performed at the Phase I Unit for study by the 1st screened subject. The last subject last visit (LSLV) is defined as the last visit performed at the Phase I Unit by the last subject in study, i.e., the last visit foreseen by the study protocol, independently of the fact that the subject is a completer or a withdrawn subject.

The following phases, visits and procedures are performed:

#### > Screening phase

- Screening visit 1: between Day -21 and Day -2
- Visit 2: Day -1

#### > Interventional phase

■ Visit 3: Days 1-2

#### > Final phase

• Visit 4: Day 7: Final visit or Early termination visit (ETV). In case of early discontinuation, discontinued subjects will undergo an ETV.



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Screening – visit 1 | From Day -21 to<br>Day -2 | <ul> <li>Explanation to the subject of study aims, procedures and possible risks</li> <li>Informed consent signature</li> <li>Screening number assignment (as S001, S002, etc.)</li> <li>Demographic data and lifestyle recording</li> <li>Medical/surgical history</li> <li>Previous/concomitant medications</li> <li>Full physical examination (body weight, height, body mass index, vital signs, physical abnormalities)</li> <li>Triplicate 12-lead ECG recording</li> <li>Laboratory analyses: hematology, blood chemistry, urinalysis and virology</li> <li>Serum pregnancy test (women only)</li> <li>Urine multi-drug screening test</li> <li>AE recording</li> <li>Inclusion/exclusion criteria evaluation</li> </ul> | Note: The first two letters of the surname followed by the first two letters of the first name will be used in the Phase I Unit source document only and will not be transferred to the Sponsor |
| Visit 2 | Day -1 | <ul> <li>Short physical examination (only if screening physical examination performed more than 7 days before Day -1)</li> <li>Recording of concomitant medications</li> <li>Salivary alcohol test</li> <li>Urine pregnancy test (women only)</li> <li>Urine multi-drug screening test</li> <li>Body weight</li> <li>Vital signs measurement</li> <li>AE recording</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Eligibility evaluation</li> <li>Enrolment</li> <li>Subject study number assignment (as 001, 002, etc.)</li> </ul> | Arrival at the Phase I Unit in the evening Confinement until the morning of Day 2 Standardized low-fat dinner Fasting for 10 h (overnight) |
| Visit 3 | Day 1 | <ul> <li>T or Rα treatment</li> <li>Vital signs measurement</li> <li>Triplicate 12-lead ECG recording</li> <li>Blood sample collection for PK analysis</li> <li>Recording of concomitant medications</li> <li>AE recording</li> </ul> | Standardized lunch at about 13:00 (5 h post-dose) Standardized dinner at about 20:00 (12 h post-dose) |
| Vis | Day 2 | <ul> <li>Vital signs measurement</li> <li>Triplicate 12-lead ECG recording</li> <li>Blood sample collection for PK analysis</li> <li>Recording of concomitant medications</li> <li>Short physical examination upon discharge</li> <li>AE recording</li> </ul> | Discharge from the Phase I Unit in the morning after the 24-h post-dose blood sample collection, ECG recording and vital signs check |



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Visit 4 - Final Visit/ETV | Day 7 /<br>at ETV in case<br>of<br>discontinuation | <ul> <li>Full physical examination (body weight and physical abnormalities)</li> <li>Recording of concomitant medications</li> <li>Vital signs measurement</li> <li>Triplicate 12-lead ECG recording</li> <li>Urine pregnancy test (women only)</li> <li>Laboratory analyses as at screening, except for virology</li> <li>AE recording</li> <li>In case of clinically significant results at the final visit, the subjects will be followed-up by the Investigator until the normalization of the concerned clinical parameter(s)</li> </ul> | Upon leaving, the subjects will be instructed to contact immediately the Investigator in case of occurrence of any adverse reactions |



# 5.2 Decisional process for escalation to next administration duration

All TEAEs will be recorded in the CRF. TEAEs will be assessed by the Investigator with focus on general safety and local tolerability (i.e., any TEAEs appearing after start of injection and interesting the injection arm).

Following all planned subject's safety assessments and before subject's discharge, the Investigator will evaluate the reported TEAEs.

#### 5.2.1 Decisional process for treatment of subjects within the cohorts

Subjects belonging to cohort 2, 3 and 4 will be sequentially treated as 3 subgroups of 3, 3 and 4 subjects respectively, in each cohort.

Following the treatment of the first 3 subjects in the cohort, the collected safety parameters will be carefully assessed by the Investigator. In particular, the local tolerability will be evaluated in view of confirming the treatment of the next subgroup of 3 subjects in the same cohort.

If deemed necessary, the study Investigator will contact the Sponsor Medical Expert and seek advice.

The same process will be repeated following the second subgroup of 3 subjects for confirming the treatment of the last 4 subjects of the cohort.

#### 5.2.2 Decisional process for escalation to next administration duration

Following the completion of each cohort, the Sponsor Medical Expert will be provided with a summary of the observed tolerability, detailing each TEAE reported up to 60 min after the end of infusion of T and up to subject's discharge on Day 2. The Investigator will provide his assessments on severity and relationship to T. The Investigator will also provide a conclusion on the systemic and local tolerability related to the administration duration of T tested in the cohort, including his suggestion whether to consider safe to proceed with treating the next cohort of subjects with the next predefined infusion duration of T.

If the safety data obtained from a T treated cohort are considered as not sufficient for taking a decision on the infusion duration de-escalation process, and if additional safety data are deemed necessary to allow such decision to be taken, the study Investigator and the Sponsor Medical Expert may decide to add additional subjects (up to a maximum of 4 subjects per cohort) to the 10 subjects of the treated cohort.

The Sponsor Medical Expert will confirm the Sponsor's agreement to proceed or not with the treatment of the next planned subjects' cohort / injection duration.

Study will be stopped if any of the following criteria is met:

- 1. Any serious adverse event (SAE) assessed as at least possibly related to T experienced within 60 min after the end of T injection by at least one subject in a cohort.
- 2. Any AE coded with the same preferred term (PT) occurring to 2 subjects of the same cohort with both AEs judged at least as possibly related to T and of severe intensity, within 60 min after the end of T injection.



3. Any AE coded with the same PT occurring to 3 (or more) subjects of the same cohort with the AEs judged at least as possibly related to T and of moderate intensity, within 60 min after the end of T injection.

#### 5.3 Diet and lifestyle

During the subjects' confinement at the Phase I Unit, they will not take any food or drinks (except water) for about 10 h (i.e., overnight) before P, T or R. Water will be allowed as desired, except for 1 h before and 1 h after P, T or R administration start. In order to maintain an adequate hydration, the subjects will be encouraged to drink at least 180 mL of still mineral water every 2 h for 5 h post-dose, starting at 1 h post-dose.

On Day 1 the subjects will remain fasted until 5 h after the start of injection/infusion. Standardized lunch and dinner will be served at approximately 5 h and 12 h after the start of injection/infusion.

On Day -1 a standardized low-fat dinner will be served. One cup of coffee or tea will be allowed after each meal only; any other coffee, tea or food containing xanthines (i.e., coke, energy drinks, chocolate, etc.), alcohol and grapefruit will be forbidden during confinement. In particular, grapefruit and any other food or beverage known to interfere with cytochrome P450 will be forbidden for 7 days (168 h) before the first study treatment administration until the end of the study.

During confinements, smoking will be forbidden.

During confinement, routine ambulant daily activities will be strongly recommended.

#### 5.4 Restrictions

The subjects will be confined from the evening preceding T or  $R\alpha$  (undiluted R) treatment (study Day -1) until the morning of Day 2. All other study visits will be ambulatory. During confinement, hazardous, strenuous or athletic activities will not be permitted.



# 6 STUDY SUBJECT IDENTIFICATION METHOD AND TREATMENT ASSIGNMENT METHOD

# 6.1 Unique subject identifier

All the subjects who sign the informed consent form for each part of the present study will be coded with "unique subject identifiers" when data are extracted from the study database into the domains of the CDISC SDTM model.

The unique subject identifier consists of the sponsor study code (i.e., PNET-22-08), the 3-digit site number (i.e., 001), the 4-digit screening number (e.g., S001, S002, etc.) and, if applicable, the 3-digit subject study number (e.g., 001, 002, etc.). Study code, site number, screening number and subject study or randomization number are separated by slashes ("/").

# 6.2 Subject identifier for the study

The last 8 digits of the unique subject identifier (enrolled subjects), corresponding to the subject screening and subject study numbers separated by a slash, or the last 4 digits of the unique subject identifier (not enrolled subjects), corresponding to the subject screening number, will appear as subject identifier in the individual listings and figures of the clinical study report and will be used to identify the subjects in in-text tables or wording (if applicable).

#### 6.3 Randomisation

Cohorts are not randomized.

#### 6.4 Treatment allocation

In cohort 1, the subjects will be assigned to one parallel treatment (T or  $R\alpha$ ) according to their admittance to the Phase I Unit, i.e., the first 10 subjects will receive  $R\alpha$  and the next ten T.

#### 6.5 Blinding

This is an open-label study. No masking procedure will be applied.



#### 7 STUDY EVALUATION PARAMETERS

#### 7.1 Study variables

#### 7.1.1 Primary safety variables

• Type, number and frequency of TEAEs collected up to 24 h post-dose.

## 7.1.2 Secondary safety variables

The assessment of safety and tolerability of the IMP is based on treatment-emergent adverse events, vital signs (blood pressure and pulse rate), 12-lead ECG, clinical laboratory tests (blood chemistry, hematology and urinalysis), body weight and physical examination.

# 7.2 PK parameters

For plasma fosnetupitant, netupitant and its main metabolites M1, M2 and M3, when applicable, the following parameters will be measured/calculated:

- C<sub>0</sub>: Plasma concentration at the end of the injection or infusion
- C<sub>max</sub>: Maximum concentration
- $t_{max}$ : Time to achieve  $C_{max}$
- C<sub>last</sub>: Last measurable plasma concentration above the lower limit of quantification of the bioanalytical method
- t<sub>last</sub>: Time of last measurable plasma concentration above the lower limit of quantification of the bioanalytical method
- AUC<sub>0-t</sub>: Area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method
- AUC<sub>0-24</sub>: Area Under the concentration-time Curve from time zero to 24h
- $\lambda_z$ : Terminal elimination rate constant, calculated, if feasible, by log-linear regression using at least 3 points, C<sub>0</sub> and C<sub>max</sub> excluded
- t<sub>1/2</sub>: Apparent terminal half-life, calculated, if feasible, as  $ln2/\lambda_z$
- CL: Systemic clearance
- Vz: Apparent volume of distribution in the post-distribution phase
- MRT: Mean residence time

The quality of log-linear regression (and, consequently, the reliability of the extrapolated PK parameters) should be demonstrated by a determination coefficient  $R_2 \ge 0.8$ . Individual extrapolated parameters, when considered unreliable, will be reported as NC (not calculated).



#### 8 STATISTICAL METHOD

The data documented in this study and the parameters measured will be evaluated and compared using classic descriptive statistics, i.e., geometric mean (PK data only), arithmetic mean, SD, CV (%), minimum, median and maximum values for quantitative variables, and frequencies for qualitative variables.

Not available data are evaluated as "missing values". The statistical analysis of demographic and safety data is performed using SAS® version 9.3 (TS1M1) (8) or higher (the actual version is stated in the final report).

The statistical analysis of PK parameters is performed using Phoenix WinNonlin® version 8.3.5 (9) or higher and SAS® version 9.3 (TS1M1) or higher.

Demographic, safety, and PK analyses will be performed by the Biometry Unit of the CRO, while ECG statistical analysis will be performed by the provider of continuous ECG.

# 8.1 Tables, listings and figures layout

Tables, listings and figures are provided according to the following settings:

- Background: White
- Foreground: Black
- Font face: Times
- Font style: Roman
- Font size: 10 pt
- Font weight: Medium (data, footers and notes), Bold (titles and headers)
- Font width: Normal
- Layout: Landscape
- Top Margin: 2.5 cm
- Bottom Margin: 2.5 cm
- Left Margin: 0.8 cm
- Right Margin: 0.8 cm
- Test label: T
- Reference label: Rα
- Cohort label: Cohort 1 30 min (Rα), Cohort 1 30 min (T), Cohort 2 15 min (T), Cohort 3 5 min (T), Cohort 4 2 min (T)
- Date format: ddMMMyyyy
- Means, standard deviations, percent coefficient of variations, medians, lower confidence limits and upper confidence limits are rounded to one digit more than the original data
- Minima and maxima keep the same number of decimal digits as the source values
- p-values are rounded to the fourth decimal digit and are flagged by an asterisk (\*) in case of statistical significance (i.e. p-value < 0.05 or, in case of centre by treatment interaction, p-value < 0.10)
- p-values lower than 0.0001 are reported as "<.0001 \*".

Data and results will be presented by cohort to which the subject belongs. For Cohort 1 data will be presented separately for subjects who received reference or test product.



#### 8.2 Analysis sets

#### 8.2.1 Definitions

A subject will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A subject will be defined as <u>eligible</u> if he/she meets all the inclusion/exclusion criteria. Otherwise, he/she will be defined as a screen failure.

A subject will be defined as <u>enrolled</u> in the study if he/she is included in the interventional phase of the study. The enrolment will be performed through a non-randomized inclusion in the study.

An eligible but not enrolled subject will be defined as a reserve.

The following analysis sets are defined:

- *Enrolled set*: all enrolled subjects. This analysis set will be used for demographic, baseline and background characteristics
- Safety set: all subjects who receive at least one dose of the IMPs, including partial administration. This analysis set will be used for the safety analyses
- *PK set*: all enrolled subjects who fulfil the study protocol requirements in terms of T or Rα administration and have evaluable PK data readouts, with no major deviations that may affect the PK results. This analysis set will be used for the statistical analysis of the PK results.

Each subject will be coded by the CRO Biometry Unit as valid or not valid for the Safety set, PK set. Subjects will be evaluated according to the treatment they actually receive.

#### 8.2.2 Reasons for exclusion from the PK Set

Reasons for the exclusion of subjects from one period in the PK set are the following:

- intake of concomitant medications or food / beverages which could render the plasma concentration-time profile unreliable
- AEs which could render the plasma concentration-time profile unreliable
- administration errors which could render the plasma concentration-time profile unreliable
- > other events which could render the plasma concentration-time profile unreliable

If one of these events occurs, it will be noted in the CRF as the study is being conducted.

#### 8.3 Sample size and power considerations

The planned number of 20 healthy subjects to be included in cohort 1 and of 10 healthy subjects to be included in each following cohort (cohorts 2, 3 and 4) of the study was not computed by statistical assumptions.



# 8.4 Demographic, baseline and background characteristics

Critical demographic characteristics will be examined according to qualitative or quantitative data. Qualitative data will be summarized in contingency tables. Quantitative data will be summarized using classic descriptive statistics.

## 8.4.1 Subjects' disposition

The disposition of all subjects enrolled in the study will be listed (Listing 16.2.4.1) and summarised by cohort and overall (Table 14.1.1.1). The number and proportion of subjects enrolled, treated and completing the study, the number and proportion of withdrawals and the reasons for withdrawal will be presented.

# 8.4.2 Analysis sets

The subjects included in each analysis sets will be summarised by cohort and overall (Table 14.1.1.2).

# 8.4.3 Subjects excluded from PK and/or safety analysis

All subjects excluded from the PK and/or safety analysis will be listed and the reasons for exclusion will be reported (Listing 16.2.3.1).

#### 8.4.4 Discontinued subjects

All subjects who discontinued the clinical trial (if any) will be listed (Listing 16.2.1.1). Last IMP administered before discontinuation, gender, age, last visit performed before discontinuation, time elapsed from last IMP administration (hours), date of premature discontinuation and primary reason for subject premature discontinuation will be reported.

#### 8.4.5 Protocol deviations

All the protocol deviations reported during the clinical trial will be listed (Listing 16.2.2.1) and summarised by cohort and overall classified as minor and major (Table 14.1.1.5). The number and proportion of subjects for each deviation will be reported.

#### 8.4.6 Demography

Demographic data will be listed (Listing 16.2.4.2) and summarised by cohort and overall (Table 14.1.1.3). The number and proportion of subjects in each category for categorical variables (sex and race) and descriptive statistics (mean, SD, CV%, minimum, median and maximum) for continuous variables (age, body weight, height, BMI) will be presented.

#### 8.4.7 Physical examination

Date of the physical examination at screening, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.4.4).



#### 8.4.8 Fertility status and contraceptive method

The fertility status and the contraceptive method used by the female subjects will be listed (Listing 16.2.10.6).

## 8.4.9 Reproductive status and contraception

The reproductive status and the contraceptive method used by the male subjects will be listed (Listing 16.2.10.7).

# 8.4.10 Salivary alcohol test, pregnancy test and urine drug test

The date/time of the result of salivary alcohol test, pregnancy test and urine drug test will be listed (Listing 16.2.8.1).

#### 8.4.11 Inclusion/exclusion criteria not met

All the unmet inclusion/exclusion criteria will be listed (Listing 16.2.4.3) and summarised by cohort and overall (Table 14.1.1.4).

#### 8.4.12 Medical and surgical history

All the diseases of medical history and the surgeries of all subjects enrolled in the study will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 27.0. and listed (Listing 16.2.10.1).

#### 8.4.13 Prior and concomitant medication

All prior and concomitant medications will be coded using the World Health Organization Drug Dictionary Enhanced (WHODDE) version March 1, 2024 and listed (Listing 16.2.10.3).

#### 8.4.14 Tobacco, alcohol and caffeine consumption

Individual tobacco, alcohol and caffeine consumption habits history collected at screening will be listed (Listing 16.2.10.4).

#### 8.4.15 Subjects' study visits

The dates of all subjects study visits will be listed (Listing 16.2.10.5).

#### **8.4.16** Meals

The date/time of the standardised meals will be listed (Listing 16.2.10.8).

#### 8.5 IMP administration

# 8.5.1 IMP administration (date/time)



The date and time of all IMP administrations and the details of the study drug interruption will be listed (Listing 16.2.5.1).

# 8.5.2 Fasting condition

The start date/time of fasting conditions and its duration will be listed (Listing 16.2.5.2).

## 8.5.3 Dose per body weight

The dose per body weight of IMP will be listed (Listing 16.2.5.3) and summarised using descriptive statistics (Table 14.3.5.6). The body weight collected at the screening visit will be used for the calculation.

# 8.6 PK analysis

The PK analysis will be performed on the subjects included into the PK Set.

#### 8.6.1 PK blood samples collection

The actual date/time of PK blood samples collection will be listed (Listing 16.2.5.4).

#### 8.6.2 Descriptive pharmacokinetics

A descriptive PK will be presented. Individual subject concentrations of fosnetupitant, netupitant and its main metabolites M1, M2 and M3, when applicable, will be presented in data listings and summarized at each time-point.

The calculated PK parameters will be listed, displayed and summarised in tables and figures. Individual and mean curves (+SD at sampling times), indicating inter-subject variability, will be plotted. Data below the lower quantification limit (BLQL) will be considered as 0 in the calculations and presented as BLQL in listings and tables. As a consequence of BLQL (i.e. 0) values, calculated geometric means (if requested) could be null. For this reason, in the presence of any null value, the geometric mean will be reported as not calculated (NC).

For plasma concentration of each analyte, descriptive statistics (N, mean, geometric mean, SD, CV%, median, minimum and maximum) will be tabulated at each time point (Table 14.2.1.1, Table 14.2.1.2, Table 14.2.1.3, Table 14.2.1.4, Table 14.2.1.5). Individual subject concentrations will be presented in data listings (Listing 16.2.5.5, Listing 16.2.5.6, Listing 16.2.5.7, Listing 16.2.5.8. Listing 16.2.5.9). All derived PK parameters will be listed (Listing 16.2.6.1, Listing 16.2.6.2, Listing 16.2.6.3, Listing 16.2.6.4, Listing 16.2.6.5) and their descriptive statistics (N, mean, geometric mean, SD, CV%, median, minimum and maximum) summarised (Table 14.2.2.1, Table 14.2.2.2, Table 14.2.2.3, Table 14.2.2.4, Table 14.2.2.5).

#### 8.7 Safety and tolerability analysis

The safety and tolerability analysis will be performed on the subjects included into the Safety Set.

#### **8.7.1** Adverse events



Adverse events (AEs) will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA) version 27.0.

AEs will be classified as pre-treatment AEs (PTAEs) and treatment-emergent AEs (TEAEs), according to the period of occurrence, as follows:

- PTAEs: all AEs occurring before the dose of IMP and not worsening after the dose of IMP
- TEAEs: all AEs occurring or worsening after the dose of IMP

Individual PTAEs and TEAEs will be listed in subject data listings (Listing 16.2.7.1, Listing 16.2.7.2).

No summary table will be provided for PTAEs.

TEAEs will be summarized by cohort and overall.

The number and percentage of subjects with any TEAE and the number of TEAEs will be presented. (Table 14.3.1.1).

The number and percentage of subjects with any TEAE and the number of TEAEs will be presented by SOC and PT (Table 14.3.1.2).

The number and percentage of subjects with any TEAE by severity and the number of TEAEs by intensity will be presented by SOC and PT (Table 14.3.1.3).

The number and percentage of subjects with any TEAE related to the IMP and the number of TEAEs related to the IMP will be presented by SOC and PT (Table 14.3.1.4).

If applicable, serious TEAE will be summarized by SOC and PT (Table 14.3.1.5) and by relationship to IMP (Table 14.3.1.6).

All TEAEs leading to death, Serious TEAEs and all TEAEs leading to discontinuation will be listed (Table 14.3.2.1).

#### 8.7.2 Vital signs

The date/time of vital signs and body weight assessments and the values of vital signs and body weight will be listed (Listing 16.2.9.1).

A table of all the abnormal vital signs' values (Table 14.3.5.1) and a table with descriptive statistics by cohort and overall will be presented (Table 14.3.5.2).

#### 8.7.3 Body weight

The date/time of body weight assessments and the values of body weight will be listed (Listing 16.2.9.1) and summarized by cohort and overall with descriptive statistics (Table 14.3.5.3).

# 8.7.4 ECG

The date/time of 12-lead ECG recording and the values of ECG parameters will be listed, as well as the overall investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) (Listing 16.2.9.2, Listing 16.2.9.3).



A table of all the abnormal ECG parameters' values by cohort and overall will be presented (Table 14.3.5.4) and the overall Investigator's interpretation will be summarized by cohort and overall using tables of frequency (Table 14.3.5.5).

#### 8.7.5 Laboratory data

The date/time of samples collection and the values of laboratory parameters will be listed, as well as the overall investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant findings (if any) (Listing 16.2.8.1, Listing 16.2.8.2).

A table of all the abnormal values by cohort and overall will be presented (Table 14.3.4.1) and the overall Investigator's interpretation will be summarized by cohort and overall using tables of frequency (Table 14.3.4.2).

## 8.7.6 Physical examination

Date of the physical examination at Day -1, if applicable, and end of the study, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be listed (Listing 16.2.10.2).

# 8.8 Analysis datasets

Analysis datasets will be created according to the version 2.1 of the ADaM model of CDISC (10).



#### 9 REFERENCES

- 1 ICH Topic E6 (R2): Good clinical practice.
- 2 ICH Topic E9: Statistical principles for clinical trials.
- 3 Study Protocol CRO-PK-23-363. "A phase I, open label, single dose, two parts study in male and female healthy subjects to assess the safety and pharmacokinetics of Fosnetupitant 235 mg administered as IV bolus and of derived Netupitant and Netupitant metabolites". Final version 3.0, 24MAY2023
- 4 Guidance for Industry. Bioavailability Studies Submitted in NDAs or INDs General Considerations. U.S. Department of Health and Human Services. Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Apr 2022
- 5 Ottoboni T, Lauw M, K MR, Cravets M, Manhard K, Clendeninn N and B Quart. HTX-019 via 2-min injection or 30-min infusion in healthy subjects. Future Oncol. 2019;15(8):865-874
- 6 ICH Topic E 8, General Considerations for Clinical Trials, CPMP/ICH/291/95, March 1998
- 7 U.S. Department of Health and Human Services and U.S. Department of Agriculture, Nutrition and your health: 2020-2025 Dietary Guidelines
- 8 SAS/STAT® User's Guide
- 9 WinNonLin Getting Started Guide, Pharsight Corporation
- 10 CDISC Analysis Data Model Version 2.1




Statistical analysis plan CRO-PK-22-363 Sponsor code PNET-22-08 Netupitant IV infusion shortening Final version 1.0, 18JUN2024

## 10 APPENDICES

- 1. Section 14 Tables Shells
- 2. Section 16.2 Individual Subject Data Listings Shells



#### Section 14 - Tables Shells

- Table 14.1.1.1 Subjects' disposition Enrolled set
- Table 14.1.1.2 Analysis sets Enrolled set
- Table 14.1.1.3 Demography Enrolled set, Safety set and PK set
- Table 14.1.1.4 Inclusion/exclusion criteria not met Enrolled set, Safety set and PK set
- Table 14.1.1.5 Protocol deviations Enrolled set, Safety set and PK set
- Table 14.2.1.1 Fosnetupitant Concentrations (ng/mL) Summary PK set
- Table 14.2.1.2 Netupitant Concentrations (ng/mL) Summary PK set
- Table 14.2.1.3 Netupitant metabolite M1 Concentrations (ng/mL) Summary PK set
- Table 14.2.1.4 Netupitant metabolite M2 Concentrations (ng/mL) Summary PK set
- Table 14.2.1.5 Netupitant metabolite M3 Concentrations (ng/mL) Summary PK set
- Table 14.2.2.1 Plasma PK parameters Fosnetupitant PK set
- Table 14.2.2.2 Plasma PK parameters Netupitant PK set
- Table 14.2.2.3 Plasma PK parameters Netupitant metabolite M1 PK set
- Table 14.2.2.4 Plasma PK parameters Netupitant metabolite M2 PK set
- Table 14.2.2.5 Plasma PK parameters Netupitant metabolite M3 PK set
- Table 14.3.1.1 Global frequency of subjects with treatment-emergent adverse events Safety set
- Table 14.3.1.2 Subjects with treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.3 Subjects with treatment-emergent adverse events by severity, system organ class and preferred term Safety set
- Table 14.3.1.4 Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.1.5 Subjects with serious treatment-emergent adverse events by system organ class and preferred term Safety set
- Table 14.3.1.6 Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term Safety set
- Table 14.3.2.1 Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation Safety set
- Table 14.3.4.1 Abnormal laboratory values Safety set
- Table 14.3.4.2 Contingency tables of investigator's interpretation of laboratory test results Safety set
- Table 14.3.5.1 Abnormal vital signs Safety set
- Table 14.3.5.2 Descriptive statistics of vital signs Safety set
- Table 14.3.5.3 Descriptive statistics of body weight Safety set
- Table 14.3.5.4 Abnormal recorded values of ECG Safety set
- Table 14.3.5.5 Contingency tables of investigator's interpretation of ECG results Safety set
- Table 14.3.5.6 Descriptive statistics of dose per body weight Safety set

CROSS Research S.A.



Table 14.1.1.1 - Subjects' disposition - Enrolled set

| | Cohort 1<br>30 min (Rα)<br>n (%) | Cohort 1<br>30 min (T)<br>n (%) | Cohort 2<br>15 min (T)<br>n (%) | Cohort 3<br>5 min (T)<br>n (%) | Cohort 4<br>2 min (T)<br>n (%) | Overall<br>n (%) |
|---|---|---|---|---|---|---|
| Enrolled | nn | nn | nn | nn | nn | nn |
| Discontinued before treatment <sup>1</sup> | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treated <sup>1</sup> | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Completed <sup>2</sup> | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Discontinued <sup>2</sup> | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Adverse event <sup>2</sup> | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Withdrawal by subject <sup>2</sup> | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects of each disposition event are reported

Note 1:The denominator for calculating the proportions is the number of enrolled subjects overall and in each cohort

Note 2: The denominator for calculating the proportions is the number of treated subjects overall and in each cohort

Source: Listing 16.2.4.1 - Subjects' disposition

Program: Tables\k363-ds-tbl.sas

CROSS Research S.A.



#### Table 14.1.1.2 - Analysis sets - Enrolled set

| | Cohort 1<br>30 min (Rα)<br>n (%) | Cohort 1<br>30 min (T)<br>n (%) | Cohort 2<br>15 min (T)<br>n (%) | Cohort 3<br>5 min (T)<br>n (%) | Cohort 4<br>2 min (T)<br>n (%) | Overall n (%) |
|---|---|---|---|---|---|---|
| Safety Set | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: The number and the proportion of subjects included in each analysis set are reported

The denominator for calculating the proportions is the number of subjects in the enrolled set overall and in each cohort

Source: Listing 16.2.3.1 - Subjects excluded from safety and/or PK analysis

Program: Tables\k363-ds-tbl.sas

CROSS Research S.A.


# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# **Cohort 1: 30 min (Rα)**

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| | В | (0/) | | 4 | ( ) |
| Sex | Female | n (%) | nn(xx.x) | nn (xx.x) | nn(xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# **Cohort 1: 30 min (Rα)**

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | xx.x | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | xx.x | XX.X | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | xx.xx |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# **Cohort 1: 30 min (Rα)**

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | xx.xx | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | xx.xx | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (T)** 

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (T)** 

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | xx.xx | xx.xx | xx.xx |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (T)** 

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | xx.xx | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | xx.xx | XX.XX | XX.XX |
| | CV% | xx.xx | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

**Cohort 2: 15 min (T)** 

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| G. | Female | (0/) | ( | | ( |
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

**Cohort 2: 15 min (T)** 

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# $Table\ 14.1.1.3-Demography-Enrolled\ set, Safety\ set\ and\ PK\ set$

**Cohort 2: 15 min (T)** 

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 3: 5 min (T)

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 3: 5 min (T)

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | xx.xx | xx.xx | xx.xx |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 3: 5 min (T)

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | xx.x | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | XX.XX | xx.xx | XX.XX |
| | SD | xx.xx | xx.xx | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | xx.xx | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 4: 2 min (T)

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 4: 2 min (T)

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | xx | XX |
| | Median | XX.X | xx.x | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

# Cohort 4: 2 min (T)

| | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

#### Overall

| | | Statistics | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|---|
| Sex | Female | n (0/) | nn (vv v) | nn (vv v) | nn (vv v) |
| Sex | | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Ethnicity | Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not Hispanic or Latino | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Not reported | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Unknown | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age [years] | | N | nn | nn | nn |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

#### Overall

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Age [years] | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Height [cm] | N | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX |
| Body Weight [kg] | N | nn | nn | nn |
| | Mean | xx.xx | xx.xx | xx.xx |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography

Program: Tables\k363-dm-tbl.sas



# Table 14.1.1.3 - Demography - Enrolled set, Safety set and PK set

#### Overall

| | Statistics | Enrolled Set N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|---|
| Body Weight [kg] | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |
| Body Mass Index [kg/m²] | N | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X |
| | Median | XX.XX | XX.XX | XX.XX |
| | Max | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the cohort they belong to

Note 1: The number and the proportion of subjects of each sex and race are reported

Note 2: The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.3 - Demography Program: Tables\k363-dm-tbl.sas



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (Rα)** 

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

 $Program: Tables \backslash k363\text{-}ie\text{-}tbl.sas$ 



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (T)** 

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program: Tables\k363-ie-tbl.sas



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

**Cohort 2: 15 min (T)** 

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program: Tables\k363-ie-tbl.sas



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

# Cohort 3: 5 min (T)

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort \_

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program: Tables\k363-ie-tbl.sas



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

#### Cohort 4: 2 min (T)

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort \_

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program: Tables\k363-ie-tbl.sas



### Table 14.1.1.4 - Inclusion/exclusion criteria not met - Enrolled set, Safety set and PK set

# Overall

| | Enrolled Set | Safety Set | PK Set |
|---|---|---|---|
| | N=XX | N=XX | N=XX |
| Number of subjects with any inclusion/exclusion criteria not met | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 [Informed consent] Inclusion criterion 2 [Sex and Age] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 [ECG (12-leads, supine position)] Exclusion criterion 2 [Physical findings] | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any criterion not met are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program:Tables\k363-ie-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (Rα)** 

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn (xx.x) | nn(xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Medication not admitted | nn(xx.x) | nn (xx.x) | nn(xx.x) |
| <del></del> | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | nn (xx.x) | nn (xx.x) | nn(xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

**Cohort 1: 30 min (T)** 

| Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn (xx.x) | nn(xx.x) | nn(xx.x) |
| nn(xx.x) | nn(xx.x) | nn(xx.x) |
| nn(xx.x) | nn(xx.x) | nn(xx.x) |
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn (xx.x) | nn (xx.x) | nn (xx.x) |
| nn(xx.x) | nn(xx.x) | nn(xx.x) |
| nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | N=XX nn (xx.x) | N=XX N=XX nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

**Cohort 2: 15 min (T)** 

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Medication not admitted | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn(xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

#### Cohort 3: 5 min (T)

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Medication not admitted | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

#### Cohort 4: 2 min (T)

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Medication not admitted | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



### Table 14.1.1.5 - Protocol deviations - Enrolled set, Safety set and PK set

#### Overall

| | Enrolled Set<br>N=XX | Safety Set<br>N=XX | PK Set<br>N=XX |
|---|---|---|---|
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treatment deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criteria violation | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criteria violation | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| Medication not admitted | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled sampling time | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation from scheduled assessment time | nn(xx.x) | nn(xx.x) | nn (xx.x) |
| | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for any protocol violation are reported

The denominator for calculating the proportions is the number of subjects in each analysis set and cohort

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\k363-dv-tbl.sas



# Table 14.2.1.1 - Fosnetupitant Concentrations (ng/mL) Summary - PK set

# **Cohort 1: 30 min (Rα)**

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.1 - Fosnetupitant Concentrations (ng/mL) Summary - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.1 - Fosnetupitant Concentrations (ng/mL) Summary - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.1 - Fosnetupitant Concentrations (ng/mL) Summary - PK set

# Cohort 3: 5 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20 min</b> | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.1 - Fosnetupitant Concentrations (ng/mL) Summary - PK set

# Cohort 4: 2 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20</b> min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.2 - Netupitant Concentrations (ng/mL) Summary - PK set

# **Cohort 1: 30 min (Rα)**

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas


#### Table 14.2.1.2 - Netupitant Concentrations (ng/mL) Summary - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.2 - Netupitant Concentrations (ng/mL) Summary - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.2 - Netupitant Concentrations (ng/mL) Summary - PK set

#### Cohort 3: 5 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20 min</b> | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.2 - Netupitant Concentrations (ng/mL) Summary - PK set

#### Cohort 4: 2 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20</b> min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.3 - Netupitant metabolite M1 Concentrations (ng/mL) Summary - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.3 - Netupitant metabolite M1 Concentrations (ng/mL) Summary - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.3 - Netupitant metabolite M1 Concentrations (ng/mL) Summary - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | | | | | | | | | | - | | | | | | |
| N | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.3 - Netupitant metabolite M1 Concentrations (ng/mL) Summary - PK set

#### Cohort 3: 5 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20</b> min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX |
| CV% | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.3 - Netupitant metabolite M1 Concentrations (ng/mL) Summary - PK set

#### Cohort 4: 2 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20</b> min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.4 - Netupitant metabolite M2 Concentrations (ng/mL) Summary - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.4 - Netupitant metabolite M2 Concentrations (ng/mL) Summary - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



#### Table 14.2.1.4 - Netupitant metabolite M2 Concentrations (ng/mL) Summary - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.4 - Netupitant metabolite M2 Concentrations (ng/mL) Summary - PK set

#### Cohort 3: 5 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20</b> min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX |
| CV% | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.1.4 - Netupitant metabolite M2 Concentrations (ng/mL) Summary - PK set

Cohort 4: 2 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20 min</b> | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.5 - Netupitant metabolite M3 Concentrations (ng/mL) Summary - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.5 - Netupitant metabolite M3 Concentrations (ng/mL) Summary - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | | | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.5 - Netupitant metabolite M3 Concentrations (ng/mL) Summary - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.5 - Netupitant metabolite M3 Concentrations (ng/mL) Summary - PK set

#### Cohort 3: 5 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20 min</b> | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX |
| CV% | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



### Table 14.2.1.5 - Netupitant metabolite M3 Concentrations (ng/mL) Summary - PK set

#### Cohort 4: 2 min (T)

| Statistics | Pre | 2 min | 5 min | 10 min | 15 min | <b>20 min</b> | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | dose | | | | | | | | | | | | | | | |
| N | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Geo.Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Max | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

Source: Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Program: pk-analysis\k363-pc-tbl.sas



# Table 14.2.2.1 - Plasma PK parameters - Fosnetupitant - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_0$ | Clast | <b>t</b> last | <b>t</b> max | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| Geo.Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.1 - Plasma PK parameters - Fosnetupitant - PK set

**Cohort 1: 30 min (T)** 

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | <b>AUC</b> 0-24 | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to Source: Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.1 - Plasma PK parameters - Fosnetupitant - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to Source: Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.1 - Plasma PK parameters - Fosnetupitant - PK set

# Cohort 3: 5 min (T)

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | <b>AUC</b> 0-24 | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to Source: Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.1 - Plasma PK parameters - Fosnetupitant - PK set

# Cohort 4: 2 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to Source: Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.2 - Plasma PK parameters - Netupitant - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_{0}$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Geo.Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.2 - Plasma PK parameters - Netupitant - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.2 - Plasma PK parameters - Netupitant - PK set

**Cohort 2: 15 min (T)** 

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.2 - Plasma PK parameters - Netupitant - PK set

# Cohort 3: 5 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.2 - Plasma PK parameters - Netupitant - PK set

# Cohort 4: 2 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.3 - Plasma PK parameters - Netupitant metabolite M1 - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | C <sub>max</sub><br>(ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub><br>(ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-24</sub><br>(h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| N | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx |
| Geo.Mean | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| Max | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.3 - Plasma PK parameters - Netupitant metabolite M1 - PK set

**Cohort 1: 30 min (T)** 

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.3 - Plasma PK parameters - Netupitant metabolite M1 - PK set

**Cohort 2: 15 min (T)** 

| Statistics | C <sub>max</sub><br>(ng/mL) | C <sub>0</sub> | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-24</sub><br>(h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (lig/iliL) | (ng/mL) | (lig/iiiL) | (11) | (11) | (II lig/IIIL) | (II lig/IIIL) | (1/11) | (11) | (11112/11) | (IIIL) | (11) |
| N | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.3 - Plasma PK parameters - Netupitant metabolite M1 - PK set

# Cohort 3: 5 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.3 - Plasma PK parameters - Netupitant metabolite M1 - PK set

# Cohort 4: 2 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.4 - Plasma PK parameters - Netupitant metabolite M2 - PK set

### **Cohort 1: 30 min (Rα)**

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | <b>AUC</b> 0-24 | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.4 - Plasma PK parameters - Netupitant metabolite M2 - PK set

**Cohort 1: 30 min (T)** 

| Statistics | C <sub>max</sub><br>(ng/mL) | C <sub>0</sub> | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-24</sub><br>(h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (lig/iliL) | (ng/mL) | (lig/iiiL) | (11) | (11) | (II lig/IIIL) | (II lig/IIIL) | (1/11) | (11) | (11112/11) | (IIIL) | (11) |
| N | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$


# Table 14.2.2.4 - Plasma PK parameters - Netupitant metabolite M2 - PK set

**Cohort 2: 15 min (T)** 

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx |
| Geo.Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.4 - Plasma PK parameters - Netupitant metabolite M2 - PK set

# Cohort 3: 5 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.4 - Plasma PK parameters - Netupitant metabolite M2 - PK set

# Cohort 4: 2 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | tlast | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.5 - Plasma PK parameters - Netupitant metabolite M3 - PK set

# **Cohort 1: 30 min (Rα)**

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_{0}$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Geo.Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

Program: pk-analysis\k363-pp-tbl.sas



# Table 14.2.2.5 - Plasma PK parameters - Netupitant metabolite M3 - PK set

**Cohort 1: 30 min (T)** 

| Statistics | C <sub>max</sub><br>(ng/mL) | C <sub>0</sub> | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-24</sub><br>(h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (lig/iliL) | (ng/mL) | (lig/iiiL) | (11) | (11) | (II lig/IIIL) | (II lig/IIIL) | (1/11) | (11) | (11112/11) | (IIIL) | (11) |
| N | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.5 - Plasma PK parameters - Netupitant metabolite M3 - PK set

**Cohort 2: 15 min (T)** 

| Statistics | $\mathbf{C}_{max}$ | $\mathbf{C}_{0}$ | $\mathbf{C}_{last}$ | tlast | tmax | AUC <sub>0-t</sub> | <b>AUC</b> <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | xxx.xx | xxx.xx | xxx.xx |
| Geo.Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Mean | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

 $Program: pk-analysis \verb|\k363-pp-tbl.sas|$ 



# Table 14.2.2.5 - Plasma PK parameters - Netupitant metabolite M3 - PK set

# Cohort 3: 5 min (T)

| Statistics | Cmax | $\mathbf{C}_0$ | Clast | <b>t</b> last | tmax | AUC <sub>0-t</sub> | AUC <sub>0-24</sub> | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| N | xxx.xx | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| CV% | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Min | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Median | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Max | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.2.2.5 - Plasma PK parameters - Netupitant metabolite M3 - PK set

# Cohort 4: 2 min (T)

| Statistics | C <sub>max</sub><br>(ng/mL) | C <sub>0</sub> | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>0-t</sub><br>(h*ng/mL) | AUC <sub>0-24</sub><br>(h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (lig/iliL) | (ng/mL) | (lig/iiiL) | (11) | (11) | (II lig/IIIL) | (II lig/IIIL) | (1/11) | (11) | (11112/11) | (IIIL) | (11) |
| N | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| Geo.Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX |
| Mean | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| CV% | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Min | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Median | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx |
| Max | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx |

Note: Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

 $Program: pk-analysis \verb|\k| 363-pp-tbl.sas$ 



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 1: 30 min (Rα)** 

| | Safety Set N=XX n (%) [n AE] |
|-----------------------------------|----------------------------------|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | nn(xx.x)[kk] |
| Related Not related | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Severity | nn (xx.x) [kk] |
| Mild<br>Moderate | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Severe | nn (xx.x) [kk] |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 1: 30 min (Rα)** 

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | $\operatorname{nn}(xx.x)[kk]$ |
| Relationship | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |
| Related Not related | nn (xx.x) [kk] $nn (xx.x) [kk]$ |
| Severity | nn (xx.x) [kk] |
| Mild Moderate | nn(xx.x)[kk] $nn(xx.x)[kk]$ |
| Severe | nn (xx.x) [kk] |
| Leading to discontinuation | $\operatorname{nn}(xx.x)[kk]$ |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

 $Program: Tables \verb|\k363-ae-01-tbl.sas|$ 



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 1: 30 min (T)** 

| | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | $\operatorname{nn}(xx.x)[kk]$ |
| Relationship | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |
| Related Not related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | $\operatorname{nn}\left(\mathbf{x}\mathbf{x}.\mathbf{x}\right)\left[\mathbf{k}\mathbf{k}\right]$ |
| Severity | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |
| Mild | $\operatorname{nn}(xx.x)[kk]$ |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | $\operatorname{nn}(\mathbf{x}\mathbf{x}.\mathbf{x})[\mathbf{k}\mathbf{k}]$ |
| Leading to discontinuation | nn(xx.x)[kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 1: 30 min (T)** 

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | $\operatorname{nn}(xx.x)[kk]$ |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn (xx.x) [kk] |
| Severity | $\operatorname{nn}(xx.x)[kk]$ |
| Mild | nn(xx.x)[kk] |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | $\operatorname{nn}(xx.x)[kk]$ |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



## Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 2: 15 min (T)** 

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | nn(xx.x)[kk] |
| Relationship | nn(xx.x)[kk] |
| Related | $\operatorname{nn}(\mathbf{x}\mathbf{x}.\mathbf{x})[\mathbf{k}\mathbf{k}]$ |
| Not related | $\operatorname{nn}(xx.x)[kk]$ |
| Severity | $\operatorname{nn}\left(\mathbf{x}\mathbf{x}.\mathbf{x}\right)\left[\mathbf{k}\mathbf{k}\right]$ |
| Mild | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |
| Moderate | $\operatorname{nn}\left(\mathbf{x}\mathbf{x}.\mathbf{x}\right)\left[\mathbf{k}\mathbf{k}\right]$ |
| Severe | $\operatorname{nn}(xx.x)[kk]$ |
| Leading to discontinuation | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

**Cohort 2: 15 min (T)** 

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | $\operatorname{nn}(xx.x)[kk]$ |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn (xx.x) [kk] |
| Severity | $\operatorname{nn}(xx.x)[kk]$ |
| Mild | nn(xx.x)[kk] |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | $\operatorname{nn}(xx.x)[kk]$ |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

# Cohort 3: 5 min (T)

| | Safety Set N=XX n (%) [n AE] |
|-----------------------------------|----------------------------------|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | nn (xx.x) [kk] |
| Related Not related | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Severity | nn (xx.x) [kk] |
| Mild<br>Moderate | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| Severe | nn (xx.x) [kk] |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

## Cohort 3: 5 min (T)

| | Safety Set N=XX n (%) [n AE] |
|-------------------------------------------|-------------------------------|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | nn (xx.x) [kk] |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn(xx.x)[kk] |
| Severity | nn (xx.x) [kk] |
| Mild | nn(xx.x)[kk] |
| Moderate | nn(xx.x)[kk] |
| Severe | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

## Cohort 4: 2 min (T)

| | Safety Set N=XX n (%) [n AE] |
|-----------------------------------|-------------------------------|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | $\operatorname{nn}(xx.x)[kk]$ |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn (xx.x) [kk] |
| Severity | nn (xx.x) [kk] |
| Mild | $\operatorname{nn}(xx.x)[kk]$ |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

## Cohort 4: 2 min (T)

| | Safety Set N=XX n (%) [n AE] |
|-------------------------------------------|-------------------------------|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | nn (xx.x) [kk] |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn(xx.x)[kk] |
| Severity | nn (xx.x) [kk] |
| Mild | nn(xx.x)[kk] |
| Moderate | nn(xx.x)[kk] |
| Severe | nn(xx.x)[kk] |
| Leading to discontinuation | nn(xx.x)[kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



# Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

#### Overall

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | nn(xx.x)[kk] |
| Related Not related | nn (xx.x) [kk] $nn (xx.x) [kk]$ |
| Severity Mild | $\operatorname{nn}(xx.x)[kk]$ $\operatorname{nn}(xx.x)[kk]$ |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | $\operatorname{nn}(xx.x)[kk]$ |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



## Table 14.3.1.1 - Global frequency of subjects with treatment-emergent adverse events - Safety set

#### Overall

| | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Relationship | $\operatorname{nn}(xx.x)[kk]$ |
| Related | $\operatorname{nn}(xx.x)[kk]$ |
| Not related | nn (xx.x) [kk] |
| Severity | $\operatorname{nn}(xx.x)[kk]$ |
| Mild | nn(xx.x)[kk] |
| Moderate | $\operatorname{nn}(xx.x)[kk]$ |
| Severe | $\operatorname{nn}(xx.x)[kk]$ |
| Leading to discontinuation | nn (xx.x) [kk] |

Note: Subjects are summarised according to the relationship and severity reported

The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported

The denominator for calculating the proportions is the number of subjects in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-01-tbl.sas



## Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 1: 30 min (Rα)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | nn(xx.x)[kk] |
| Nervous system disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Headache | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper<br>Diarrhoea | $\begin{array}{c} nn \ (xx.x) \ [kk] \\ nn \ (xx.x) \ [kk] \end{array}$ |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 1: 30 min (T)** 

| Safety Set |
|----------------|
| N=XX |
| n (%) [n AE] |
| nn (xx.x) [kk] |
| nn (xx.x) [kk] |
| nn (xx.x) [kk] |
| <b></b> |
| nn(xx.x)[kk] |
| nn (xx.x) [kk] |
| nn (xx.x) [kk] |
| <b></b> |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 2: 15 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Nervous system disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Headache | nn (xx.x) [kk] |
| ••• | |
| Gastrointestinal disorders | $\operatorname{nn}(\mathbf{x}\mathbf{x}.\mathbf{x})[\mathbf{k}\mathbf{k}]$ |
| Abdominal pain upper | $\operatorname{nn}(xx.x)[kk]$ |
| Diarrhoea | nn (xx.x) [kk]<br> |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

## Cohort 3: 5 min (T)

| | Safety Set |
|-----------------------------------|----------------------------------------|
| System Organ Class <sup>1</sup> | N=XX |
| Preferred Term <sup>1</sup> | n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(xx.x)[kk] |
| | \ /L ] |
| Nervous system disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Tel Foul by stelli diborders | mr (MMA) [MK] |
| Headache | $\operatorname{nn}(xx.x)[kk]$ |
| Heddache | $\min (\lambda \lambda, \lambda) [KK]$ |
| ··· | ··· |
| | ( ) [II] |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper | $\operatorname{nn}(xx.x)[kk]$ |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

## Cohort 4: 2 min (T)

| | Safety Set |
|-----------------------------------|----------------------------------------|
| System Organ Class <sup>1</sup> | N=XX |
| Preferred Term <sup>1</sup> | n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(xx.x)[kk] |
| | \ /L ] |
| Nervous system disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Tel Foul by stelli diborders | mr (MMA) [MK] |
| Headache | $\operatorname{nn}(xx.x)[kk]$ |
| Heddache | $\min (\lambda \lambda, \lambda) [KK]$ |
| ··· | ··· |
| | ( ) [II] |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper | $\operatorname{nn}(xx.x)[kk]$ |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.2 - Subjects with treatment-emergent adverse events by system organ class and preferred term - Safety set

#### Overall

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn (xx.x) [kk] |
| ··· | <b></b> |
| Gastrointestinal disorders | nn(xx.x)[kk] |
| Abdominal pain upper | nn (xx.x) [kk] |
| Diarrhoea | nn (xx.x) [kk] |
| | ··· |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

**Cohort 1: 30 min (Rα)** 

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| ··· | <b></b> | <b></b> | ··· |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas




# Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

**Cohort 1: 30 min (T)** 

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn (x.x) [kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | ··· | <b></b> | ··· |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | | <b></b> | |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

**Cohort 2: 15 min (T)** 

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn (x.x) [kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | ··· | <b></b> | ··· |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | | <b></b> | |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

## Cohort 3: 5 min (T)

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| ··· | ··· | <b></b> | <b></b> |
| Gastrointestinal disorders | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

## Cohort 4: 2 min (T)

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | | | <b></b> |
| Gastrointestinal disorders | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| Abdominal pain upper | nn (x.x) [kk] | nn (x.x) [kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



Table 14.3.1.3 - Subjects with treatment-emergent adverse events by severity, system organ class and preferred term - Safety set

#### Overall

| | | Safety Set | |
|---|---|---|---|
| System Organ Class <sup>1</sup><br>Preferred Term <sup>1</sup> | Mild<br>n (%) [n AE] | Moderate<br>n (%) [n AE] | Severe<br>n (%) [n AE] |
| Treatment-emergent Adverse Events | nn(x.x)[kk] | $\operatorname{nn}(x.x)[kk]$ | nn(x.x)[kk] |
| Nervous system disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Headache | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| ··· | <del></del> | ··· | <b></b> |
| Gastrointestinal disorders | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Abdominal pain upper | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| Diarrhoea | nn(x.x)[kk] | nn(x.x)[kk] | nn(x.x)[kk] |
| | | | <b></b> |

Note: The number and the proportion of subjects with any adverse event and the number of adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

**Cohort 1: 30 min (Rα)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| - Treferred Termi | II (70) [II AL] |
| Treatment-emergent Adverse Events related to the IMP | $\operatorname{nn}(xx.x)[kk]$ |
| Nervous system disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Headache | nn(xx.x)[kk] |
| ··· | ··· |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper | $\operatorname{nn}(xx.x)[kk]$ |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| <u></u> | |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

**Cohort 1: 30 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| | n (/v) [n 112] |
| Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper | nn(xx.x)[kk] |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| <del></del> | |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

**Cohort 2: 15 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| | n (/v) [n 112] |
| Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper | nn(xx.x)[kk] |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| <del></del> | |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

## Cohort 3: 5 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}\left(\mathbf{x}\mathbf{x}.\mathbf{x}\right)\left[\mathbf{k}\mathbf{k}\right]$ |
| Abdominal pain upper | nn (xx.x) [kk] |
| Diarrhoea | nn (xx.x) [kk] |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas


## Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

## Cohort 4: 2 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}\left(\mathbf{x}\mathbf{x}.\mathbf{x}\right)\left[\mathbf{k}\mathbf{k}\right]$ |
| Abdominal pain upper | nn (xx.x) [kk] |
| Diarrhoea | nn (xx.x) [kk] |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.4 - Subjects with treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

#### Overall

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn (xx.x) [kk] |
| Gastrointestinal disorders | <br>nn (xx.x) [kk] |
| Abdominal pain upper | nn (xx.x) [kk] |
| Diarrhoea Diarrhoea | nn(xx.x)[kk] $nn(xx.x)[kk]$ |
| | ••• |

Note: The number and the proportion of subjects with any related adverse event and the number of related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set \_

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 1: 30 min (Rα)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn(xx.x)[kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn (xx.x) [kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk]<br> |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 1: 30 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | $\operatorname{nn}(xx.x)[kk]$ |
| ··· | ••• |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper | nn(xx.x)[kk] |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| | <b></b> |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

**Cohort 2: 15 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] |
| ··· | ··· |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper | nn(xx.x)[kk] |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| | <b></b> |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

## Cohort 3: 5 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | $\operatorname{nn}(xx.x)[kk]$ |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper Diarrhoea | nn(xx.x)[kk] $nn(xx.x)[kk]$ |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

## Cohort 4: 2 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | $\operatorname{nn}(xx.x)[kk]$ |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper Diarrhoea | nn(xx.x)[kk] $nn(xx.x)[kk]$ |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.5 - Subjects with serious treatment-emergent adverse events by system organ class and preferred term - Safety set

#### Overall

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | $\operatorname{nn}(xx.x)[kk]$ |
| ··· | ••• |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper | nn(xx.x)[kk] |
| Diarrhoea | $\operatorname{nn}(xx.x)[kk]$ |
| | <b></b> |

Note: The number and the proportion of subjects with any serious adverse event and the number of serious adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set \_

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

**Cohort 1: 30 min (Rα)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set N=XX n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn(xx.x)[kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| Gastrointestinal disorders | <br>(111.1) |
| | $\operatorname{nn}\left( xx.x\right) \left[ kk\right]$ |
| Abdominal pain upper Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

**Cohort 1: 30 min (T)** 

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| <del></del> | |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

## **Cohort 2: 15 min (T)**

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| <del></del> | |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

## Cohort 3: 5 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| <del></del> | |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

## Cohort 4: 2 min (T)

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn(xx.x)[kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | <del></del> |
| Gastrointestinal disorders | $\operatorname{nn}(xx.x)[kk]$ |
| Abdominal pain upper<br>Diarrhoea | nn (xx.x) [kk]<br>nn (xx.x) [kk] |
| <del></del> | |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set \_

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



# Table 14.3.1.6 - Subjects with serious treatment-emergent adverse events related to the IMP by system organ class and preferred term - Safety set

#### Overall

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Safety Set<br>N=XX<br>n (%) [n AE] |
|---|---|
| Serious Treatment-emergent Adverse Events related to the IMP | nn (xx.x) [kk] |
| Nervous system disorders | nn (xx.x) [kk] |
| Headache | nn(xx.x)[kk] |
| <del></del> | |
| Gastrointestinal disorders | nn (xx.x) [kk] |
| Abdominal pain upper | $\operatorname{nn}(\mathbf{x}\mathbf{x}.\mathbf{x})[\mathbf{k}\mathbf{k}]$ |
| Diarrhoea | nn (xx.x) [kk] |

Note: The number and the proportion of subjects with any serious related adverse event and the number of serious related adverse events for each classification level are reported. The denominator for calculating the proportions is the number of subjects in the safety set

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-02-tbl.sas



## Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation - Safety set

# **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Adverse<br>Event | | |
|---|---|---|---|
| | ID | | |
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-03-tbl.sas



## Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation - Safety set

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Adverse<br>Event | | |
|---|---|---|---|
| | ID | | |
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-03-tbl.sas



## Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation - Safety set

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | ••• | | |

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-03-tbl.sas



## Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation - Safety set

# Cohort 3: 5 min (T)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | | | <b></b> |

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-03-tbl.sas



## Table 14.3.2.1 - Treatment-emergent adverse events leading to death, serious adverse events or treatment-emergent adverse events leading to discontinuation - Safety set

Cohort 4: 2 min (T)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | ••• | | |

Note 1: MedDRA version 27.0

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\k363-ae-03-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| <br>S001/001 | <br>End of Study | <br>ddMMMyyyy hh:mm | <br>Phosphate [mmol/L] | <br>0.84 [A] | <br>0.87 - 1.45 | <br>NCS |
| ••• | | | ··· | | ••• | |

Note: Subjects are summarised according to the cohort they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| <br>S001/001 | <br>End of Study | <br>ddMMMyyyy hh:mm | <br>Leukocytes [10^9/L] | <br>10.02 [A] | <br>4.00 - 10.00 | <br>NCS |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| <br>S001/001 | <br>End of Study | <br>ddMMMyyyy hh:mm | <br>Urinary Hemoglobin | <br>+++ [A] | <br>Absent | <br>NCS |
| ••• | | | | | | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Different from reference value

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| ••• | ••• | ••• | ••• | ••• | | ••• |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| | | | | | | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| ••• | | | | ••• | | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| | | | ··· | | ••• | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Different from reference value

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S025/023 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S025/023 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| | | | <b></b> | | | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S025/023 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S025/023 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| | | | | | ••• | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S025/023 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| | ••• | ···· | ··· | ••• | ••• | ••• |
| S025/023 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| | | | <b></b> | | ••• | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Different from reference value

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/032 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| | | | | ••• | | |
| S036/032 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| | | | | ••• | | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/032 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S036/032 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| | | | | | | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/032 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| ••• | ••• | <b></b> | <b></b> | | ••• | ••• |
| S036/032 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| ••• | ••• | | ••• | | ••• | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Different from reference value

Note 2: NCS=Not clinically significant, CS= Clinically Significant \_

Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S044/040 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S044/040 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| | | | | ••• | | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S044/040 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• |
| S044/040 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| | | | ··· | | ••• | |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Abnormal

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



# Table 14.3.4.1 - Abnormal laboratory values - Safety set

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S044/040 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S044/040 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| ••• | ••• | ••• | ••• | | | ••• |

Note: Subjects are summarised according to the group they belong to

Note 1: A=Different from reference value

Note 2: NCS=Not clinically significant, CS= Clinically Significant Source: Listing 16.2.8.1 - Individual laboratory measurements

Program: Tables\k363-lb-tbl.sas



## Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

# **Cohort 1: 30 min (Rα)**

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Program: Tables\k363-lb-tbl.sas



## Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

**Cohort 1: 30 min (T)** 

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

 $Program: Tables \verb|\k363-lb-tbl.sas|$


#### Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

**Cohort 2: 15 min (T)** 

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to \_

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



#### Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

#### Cohort 3: 5 min (T)

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to \_

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



#### Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

#### Cohort 4: 2 min (T)

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to \_

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 




#### Table 14.3.4.2 - Contingency tables of investigator's interpretation of laboratory test results - Safety set

#### Overall

| Time Point | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|
| Screening | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the group they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

 $Program: Tables \verb|\k363-lb-tbl.sas|$ 



#### Table 14.3.5.1 - Abnormal vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | NCS |
| S001/001 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 89 [L] | 100-139 | NCS |
| | | <b></b> | | | ••• | |

Note: Subjects are summarised according to the cohort they belong to

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Note 2: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k363-vs-tbl.sas



#### Table 14.3.5.1 - Abnormal vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | NCS |
| S012/011 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 89 [L] | 100-139 | NCS |
| | ••• | | <b></b> | | | ••• |

Note: Subjects are summarised according to the cohort they belong to

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Note 2: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.1 - Vital signs and body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



#### Table 14.3.5.1 - Abnormal vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S025/023 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | NCS |
| S025/023 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 89 [L] | 100-139 | NCS |
| | | | ··· | | ••• | ••• |

Note: Subjects are summarised according to the cohort they belong to

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Note 2: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k363-vs-tbl.sas



#### Table 14.3.5.1 - Abnormal vital signs - Safety set

#### Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/032 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | NCS |
| S036/032 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 89 [L] | 100-139 | NCS |
| | ••• | ··· | ··· | | ••• | ••• |

Note: Subjects are summarised according to the cohort they belong to

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Note 2: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k363-vs-tbl.sas



#### Table 14.3.5.1 - Abnormal vital signs - Safety set

#### Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S044/040 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 | NCS |
| S044/040 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 89 [L] | 100-139 | NCS |
| ••• | ••• | ··· | ··· | | ••• | ••• |

Note: Subjects are summarised according to the cohort they belong to

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Note 2: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.1 - Vital signs and body weight

Program: Tables\k363-vs-tbl.sas



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Systolic Blood Pressure [mmHg] Screening N nn Mean xxxx.x SD xxx.x CV% xxx.x Min xxx.x Median xxx.x Max xxx Systolic Blood Pressure [mmHg] Visit 2 N nn Mean xxx.x SD xxx.x SD xxx.x N Median xxx.x Median xxx.x Max xxx Systolic Blood Pressure [mmHg] N nn Mean xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x CV% xxx.x Xxx.x | Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|---|
| Mean | Systolic Blood Pressure [mmHg] | Screening | N | nn |
| SD | Systeme Brood Fressure [mmrtg] | Sereeming | | |
| CV% xxx.x Min xxx Min xxx Median xxx.x Max xxx xxx | | | | |
| Systolic Blood Pressure [mmHg] Visit 2 N Median XXX. Max N Mean XXX.X SD XXX.X CV% Min Min XXX.X Min Median XXX.X Min Median XXX.X Min Median XXX.X X Median XXX.X X SD XXX.X X SD XXX.X X Min Median XXX.X X SD XXX.X X XXX X XXX X SD XXX.X X XXX X XXX XXX X XXX X XXX X XXX X XXX X | | | | |
| Systolic Blood Pressure [mmHg] Visit 2 N Mean SSD CV% XXX.X Min Median XXX.X Min Median XXX.X Median XXX.X Median XXX.X Median XXX.X Median XXX.X Median XXX.X Median XXX.X Max XXX SD Systolic Blood Pressure [mmHg] N Mean XXX.X SD XXX.X SD XXX.X | | | | |
| Systolic Blood Pressure [mmHg] Visit 2 N Mean XXX.X SD XXX.X CV% Min XXX Median XXX.X Median XXX.X Median XXX.X Median XXX.X Max XXX SD Systolic Blood Pressure [mmHg] N Mean XXX.X SD N Mean XXX.X SD XXX.X XX | | | | |
| Mean xxx.x SD | | | | XXX |
| Mean xxx.x SD | Systolic Blood Pressure [mmHa] | Visit 2 | N | nn |
| SD | Systeme Blood Fressure [mining] | VISIC Z | | |
| CV% xxx.x Min xxx Median xxx.x Median xxx.x Max xxx.x Max xxx.x Max xxx.x Max xxx Max xxx xxx xxx Xxx Xxx Xxx Xxx Xxx Xxx X | | | | |
| Min xxx Median xxx.x Max xxx.x Max xxx.x Systolic Blood Pressure [mmHg] N nn Mean xxx.x Mean xxx.x SD xxx.x | | | | |
| Median xxx.x Max xxx Systolic Blood Pressure [mmHg] N nn Mean xxx.x Mean xxx.x SD xxx.x | | | | |
| Systolic Blood Pressure [mmHg] N nn Mean xxx.x SD xxx.x | | | | |
| Systolic Blood Pressure [mmHg] N nn Mean xxx.x SD xxx.x | | | | |
| Mean xxx.x SD xxx.x | | | | |
| Mean xxx.x SD xxx.x | Systolic Blood Pressure [mmHg] | | N | nn |
| | | | Mean | XXX.X |
| CV% xxx.x | | | SD | XXX.X |
| | | | CV% | xxx.x |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |
| - | - | Mean | xxx.x |
| | | SD | XXX.X |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### **Cohort 1: 30 min (Rα)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \verb|\k363-vs-tbl.sas|$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| , | S | Mean | xxx.x |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | Ç | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | CV% | XXX.X |
| | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



# Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|------------------------|------------|------------|--------------------|
| Heart Rate [beats/min] | Screening | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 2 | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Visit 4 - Final Visit | N | nn |
| - | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| , | S | Mean | xxx.x |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | Ç | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Parameter | Time Point | Statistics | Safety Set N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Heart Rate Deats/min Screening Mean XXX.X SD XXX.X | Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|---|
| CV% XXX.X Min | Heart Rate [beats/min] | Screening | Mean | XXX.X |
| Heart Rate [beats/min] | | | SD | xxx.x |
| Heart Rate [beats/min] Visit 2 N nn Mean xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x Min Median xxx.x SD xxx.x Median xxx.x Median xxx.x Median xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Max xxx.x SD xxx.x Xxx.x Max xxx.x Xxx.x Max xxx.x Xxx.x Max xxx.x Xxx.x Mean xxx.x Xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x SD xxx.x Xxx.x Mean xxx.x Xxx.x Min xxx.x Min xxx.x Median xxx.x Xxx.x Min xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Xxx.x Median xxx.x Xxx.x Median xxx.x Xxx.x Xxx.x Median xxx.x Xxx.x Xxx.x Xxx.x Median xxx.x Xxx.x Xxx.x Xxx.x Median xxx.x Xxx.x Xx | | | CV% | xxx.x |
| Heart Rate [beats/min] Visit 2 N nn Mean xxx.x SD xxx.x CV% xxx.x Median xxx.x Median xxx.x Max xxx Heart Rate [beats/min] N nn Mean xxx.x SD xxx.x SD xxx.x SD xxx.x CV% xxx.x Min xxx.x Median xxx.x Median xxx.x Median xxx.x | | | Min | XXX |
| Heart Rate [beats/min] | | | Median | XXX.X |
| Mean xxx.x SD xxx.x CV% xxx.x Min xxx.x Median xxx.x Median xxx.x Max xxx.x Mean xxx.x Mean xxx.x Mean xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x CV% xxx.x Min xxx Min xxx.x Median xxx.x Me | | | Max | XXX |
| Mean xxx.x SD xxx.x CV% xxx.x Min xxx.x Median xxx.x Median xxx.x Max xxx.x Mean xxx.x Mean xxx.x Mean xxx.x SD xxx.x SD xxx.x SD xxx.x SD xxx.x CV% xxx.x Min xxx Min xxx.x Median xxx.x Me | Heart Rate [beats/min] | Visit 2 | N | nn |
| CV% xxx.x Min xxx Median xxx.x Median xxx.x Max xxx | | | Mean | xxx.x |
| Min xxx Median xxx.x Median xxx.x | | | SD | xxx.x |
| Median xxx.x Max xxx | | | CV% | xxx.x |
| Heart Rate [beats/min] N nn Mean xxx.x SD xxx.x CV% xxx.x Min xxx Median xxx.x | | | Min | XXX |
| Heart Rate [beats/min] N nn Mean xxx.x SD xxx.x CV% xxx.x Min xxx Median xxx.x | | | Median | XXX.X |
| Mean xxx.x SD xxx.x CV% xxx.x Min xxx Median xxx.x | | | Max | XXX |
| Mean xxx.x SD xxx.x CV% xxx.x Min xxx Median xxx.x | Heart Rate [beats/min] | | N | nn |
| SD xxx.x CV% xxx.x Min xxx Median xxx.x | . , | | Mean | XXX.X |
| CV% xxx.x Min xxx Median xxx.x | | | | XXX.X |
| Median xxx.x | | | | XXX.X |
| | | | Min | xxx |
| Max xxx | | | Median | xxx.x |
| | | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

**Cohort 2: 15 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Visit 4 - Final Visit | N | nn |
| - | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| Systeme Blood Pressure [mmm15] | Sercening | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| [6] | 2000 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|------------------------|------------|------------|--------------------|
| Heart Rate [beats/min] | Screening | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Visit 4 - Final Visit | N | nn |
| 110020 21000 [0 0000 11111] | | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 4: 2 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| ., | 5 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 4: 2 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Median | XXX.X |
| | | Max | xxx |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| | Ç | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 4: 2 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | CV% | XXX.X |
| | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 4: 2 min (T)

| Parameter | <b>Time Point</b> | Statistics | Safety Set<br>N=XX |
|------------------------|-------------------|------------|--------------------|
| Heart Rate [beats/min] | Screening | Mean | XXX.X |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 2 | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | XXX.X |
| | | Max | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

## Cohort 4: 2 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | Screening | N | nn |
| , | S | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



## Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Systolic Blood Pressure [mmHg] | | Median | XXX.X |
| | | Max | XXX |
| Systolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Screening | N | nn |
| [6] | 2000 | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | xxx |
| Diastolic Blood Pressure [mmHg] | Visit 2 | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$


# Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Diastolic Blood Pressure [mmHg] | Visit 2 | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Diastolic Blood Pressure [mmHg] | Visit 4 - Final Visit | N | nn |
| | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | Screening | N | nn |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



# Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|------------------------|------------|------------|--------------------|
| Heart Rate [beats/min] | Screening | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | XXX.X |
| | | Min | XXX |
| | | Median | XXX.X |
| | | Max | XXX |
| Heart Rate [beats/min] | Visit 2 | N | nn |
| - | | Mean | xxx.x |
| | | SD | xxx.x |
| | | CV% | xxx.x |
| | | Min | xxx |
| | | Median | xxx.x |
| | | Max | XXX |
| Heart Rate [beats/min] | | N | nn |
| | | Mean | XXX.X |
| | | SD | XXX.X |
| | | CV% | xxx.x |
| | | Min | XXX |
| | | Median | xxx.x |
| | | Max | xxx |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program:Tables\k363-vs-tbl.sas



# Table 14.3.5.2 - Descriptive statistics of vital signs - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|---|---|---|---|
| Heart Rate [beats/min] | Visit 4 - Final Visit | N<br>Mean<br>SD<br>CV%<br>Min<br>Median | nn<br>xxx.x<br>xxx.x<br>xxx.x<br>xxx |
| | | Max | XXX |

Subjects are summarised according to the cohort they belong to

Source: Listing 16.2.9.1 - Vital signs and Body weight

 $Program: Tables \backslash k363\text{-}vs\text{-}tbl.sas$ 



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

## **Cohort 1: 30 min (Rα)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|------------|--------------------|
| Weight [kg] | Screening | N | nn |
| | | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn |
| 5 1 51 | · | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |

Note: Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|--------------|--------------|------------|--------------------|
| Weight [kg] | Screening | N | nn |
| Wording [Mg] | Sereeming | Mean | XXX.XX |
| | | SD | xxx.xx |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn. |
| weight [kg] | End of Study | | nn |
| | | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | xxx.xx |
| | | Max | xxx.x |

Note:Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

# **Cohort 2: 15 min (T)**

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|------------|--------------------|
| Waink flan | Camanina | N | |
| Weight [kg] | Screening | N | nn |
| | | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn |
| | Ž | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | xxx.xx |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |

Note:Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

# Cohort 3: 5 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|---------------|--------------------|
| Weight [kg] | Screening | N<br>Mean | nn<br>xxx.xx |
| | | SD<br>CV% | xxx.xx<br>xxx.xx |
| | | Min<br>Median | XXX.X<br>XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn |
| | | Mean<br>SD | XXX.XX<br>XXX.XX |
| | | CV%<br>Min | xxx.xx<br>xxx.x |
| | | Median | XXX.XX |
| | | Max | XXX.X |

Note:Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

# Cohort 4: 2 min (T)

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|--------------|--------------|------------|--------------------|
| Weight [kg] | Screening | N | nn |
| Wording [Mg] | Sereeming | Mean | XXX.XX |
| | | SD | xxx.xx |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn. |
| weight [kg] | End of Study | | nn |
| | | Mean | XXX.XX |
| | | SD | XXX.XX |
| | | CV% | XXX.XX |
| | | Min | XXX.X |
| | | Median | xxx.xx |
| | | Max | xxx.x |

Note:Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



# Table 14.3.5.3 - Descriptive statistics of body weight - Safety set

#### Overall

| Parameter | Time Point | Statistics | Safety Set<br>N=XX |
|-------------|--------------|---------------|--------------------|
| Weight [kg] | Screening | N<br>Mean | nn<br>xxx.xx |
| | | SD<br>CV% | xxx.xx<br>xxx.xx |
| | | Min<br>Median | XXX.X<br>XXX.XX |
| | | Max | XXX.X |
| Weight [kg] | End of Study | N | nn |
| | | Mean<br>SD | XXX.XX<br>XXX.XX |
| | | CV%<br>Min | xxx.xx<br>xxx.x |
| | | Median | XXX.XX |
| | | Max | XXX.X |

Note:Subjects are summarised according to the cohort they belong to

End of Study = Final visit or early termination visit

Source: Listing 16.2.9.1 - Vital signs and Body weight

Program: Tables\k363-vs-tbl.sas



## Table 14.3.5.4 - Abnormal recorded values of ECG - Safety set

## **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value | Clinically<br>Significant? <sup>1</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 94 | NCS |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 98 | NCS |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| | | | ••• | | ••• | |

Note: Note: Subjects are summarised according to the cohort they belong to

Note 1: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.2 - Recorded parameters of ECG, Listing 16.2.9.3 - Investigator's interpretation of ECG

Program:Tables\k363-eg-tbl.sas



## Table 14.3.5.4 - Abnormal recorded values of ECG - Safety set

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value | Clinically<br>Significant? <sup>1</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| S012/011 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 94 | NCS |
| S012/011 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 98 | NCS |
| S012/011 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| ••• | ••• | ••• | <b></b> | ···· | ••• | ••• |

Note: Note: Subjects are summarised according to the cohort they belong to

Note 1: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.2 - Recorded parameters of ECG, Listing 16.2.9.3 - Investigator's interpretation of ECG

Program:Tables\k363-eg-tbl.sas



## Table 14.3.5.4 - Abnormal recorded values of ECG - Safety set

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value | Clinically<br>Significant? <sup>1</sup> |
|---|---|---|---|---|---|---|
| S025/023 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| S025/023 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 94 | NCS |
| S025/023 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 98 | NCS |
| S025/023 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| ••• | ••• | ••• | <b></b> | ···· | ••• | ••• |

Note: Note: Subjects are summarised according to the cohort they belong to

Note 1: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.2 - Recorded parameters of ECG, Listing 16.2.9.3 - Investigator's interpretation of ECG

Program:Tables\k363-eg-tbl.sas



## Table 14.3.5.4 - Abnormal recorded values of ECG - Safety set

## Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value | Clinically<br>Significant? <sup>1</sup> |
|---|---|---|---|---|---|---|
| S036/032 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| S036/032 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 94 | NCS |
| S036/032 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 98 | NCS |
| S036/032 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| | ••• | ••• | ••• | ··· | | ••• |

Note: Note: Subjects are summarised according to the cohort they belong to

Note 1: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.2 - Recorded parameters of ECG, Listing 16.2.9.3 - Investigator's interpretation of ECG

Program:Tables\k363-eg-tbl.sas



## Table 14.3.5.4 - Abnormal recorded values of ECG - Safety set

## Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value | Clinically<br>Significant? <sup>1</sup> |
|---|---|---|---|---|---|---|
| S044/040 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| S044/040 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 94 | NCS |
| S044/040 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 98 | NCS |
| S044/040 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 96 | NCS |
| ••• | ••• | ••• | | | | |

Note: Note: Subjects are summarised according to the cohort they belong to

Note 1: NCS=Not clinically significant, CS= Clinically Significant

Source: Listing 16.2.9.2 - Recorded parameters of ECG, Listing 16.2.9.3 - Investigator's interpretation of ECG

Program:Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

## **Cohort 1: 30 min (Rα)**

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal | nn (xx.x) |
| <i>B B B B B B B B B B</i> | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| Screening | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn(xx.x) |
| Screening | 3rd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 1st | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn(xx.x) |
| End of Study | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas




#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

## **Cohort 1: 30 min (Rα)**

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

 $Program: Tables \verb|\k363-eg-tbl.sas|$ 



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

## **Cohort 1: 30 min (T)**

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal<br>Abnormal, Not Clinically Significant | nn (xx.x)<br>nn (xx.x) |
| | | Abnormal, Clinically Significant | nn(xx.x) |
| Screening | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| Screening | 3rd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 1st | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

**Cohort 1: 30 min (T)** 

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### **Cohort 2: 15 min (T)**

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| Screening | 2nd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| Screening | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | 1st | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | 2nd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

**Cohort 2: 15 min (T)** 

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### Cohort 3: 5 min (T)

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal<br>Abnormal, Not Clinically Significant | nn (xx.x)<br>nn (xx.x) |
| | | Abnormal, Clinically Significant | nn(xx.x) |
| Screening | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| Screening | 3rd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 1st | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### Cohort 3: 5 min (T)

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

 $Program: Tables \backslash k363\text{-}eg\text{-}tbl.sas$ 



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### Cohort 4: 2 min (T)

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal<br>Abnormal, Not Clinically Significant | nn (xx.x)<br>nn (xx.x) |
| | | Abnormal, Clinically Significant | nn(xx.x) |
| Screening | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| Screening | 3rd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 1st | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn (xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |
| End of Study | 2nd | Normal | nn (xx.x) |
| | | Abnormal, Not Clinically Significant | nn(xx.x) |
| | | Abnormal, Clinically Significant | nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas




#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### Cohort 4: 2 min (T)

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

 $Program: Tables \backslash k363\text{-}eg\text{-}tbl.sas$ 



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

#### Overall

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| Screening | 1st | Normal Abnormal, Not Clinically Significant Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| Screening | 2nd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| Screening | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | 1st | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |
| End of Study | 2nd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

Program: Tables\k363-eg-tbl.sas



#### Table 14.3.5.5 - Contingency tables of investigator's interpretation of ECG results - Safety set

## Overall

| Time Point | Replicate | Investigator's interpretation | Safety Set<br>N=XX |
|---|---|---|---|
| End of Study | 3rd | Normal<br>Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | nn (xx.x)<br>nn (xx.x)<br>nn (xx.x) |

Note: Subjects are summarised according to the cohort they belong to

The number and the proportion of subjects for each classification level are reported

The denominator for calculating the proportions is the number of subjects in each cohort in the safety set

Source: Listing 16.2.9.3 - Investigator's interpretation of ECG

 $Program: Tables \backslash k363\text{-}eg\text{-}tbl.sas$ 



# Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

## **Cohort 1: 30 min (Rα)**

| Parameter | Statistics | Safety Set N=XX |
|------------------------------|------------|-----------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

Program: Tables\k363-ex-tbl.sas



# Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

**Cohort 1: 30 min (T)** 

| Parameter | Statistics | Safety Set<br>N=XX |
|------------------------------|------------|--------------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

 $Program: Tables \backslash k363\text{-}ex\text{-}tbl.sas$ 



# Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

**Cohort 2: 15 min (T)** 

| Parameter | Statistics | Safety Set N=XX |
|------------------------------|------------|-----------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

Program: Tables  $\k363$ -ex-tbl.sas



# Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

# Cohort 3: 5 min (T)

| Parameter | Statistics | Safety Set<br>N=XX |
|------------------------------|------------|--------------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

Program: Tables  $\k363$ -ex-tbl.sas



## Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

## Cohort 4: 2 min (T)

| Parameter | Statistics | Safety Set N=XX |
|------------------------------|------------|-----------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

Program: Tables  $\k363$ -ex-tbl.sas



# Table 14.3.5.6 - Descriptive statistics of dose per body weight - Safety set

#### Overall

| Parameter | Statistics | Safety Set<br>N=XX |
|------------------------------|------------|--------------------|
| Dose per body weight [mg/kg] | N | nn |
| | Mean | XX.X |
| | SD | XX.X |
| | CV% | XX.X |
| | Median | XX.X |
| | Min | XX |
| | Max | XX |

Note: Subjects are summarised according to the cohort they belong to

Note: The dose per body weight was calculated using the screening body weight

Source: Listing 16.2.5.3 - Dose per body weight

Program: Tables  $\k363$ -ex-tbl.sas




Section 16.2 - Individual Subject Data Listings Shells

| Listing 16.2.1.1 - 1 | Discontinued subjects |
|----------------------|-----------------------|
|----------------------|-----------------------|

Listing 16.2.2.1 - Protocol deviations

Listing 16.2.3.1 - Subjects excluded from safety and/or PK analysis

Listing 16.2.4.1 - Subjects' disposition - Enrolled set

Listing 16.2.4.2 - Demography - Enrolled set

Listing 16.2.4.3 - Inclusion/Exclusion criteria not met - Enrolled set

Listing 16.2.4.4 - Physical examination at screening - Enrolled set

Listing 16.2.5.1 - Investigational medicinal products administration - Safety set

Listing 16.2.5.2 - Fasting conditions - Safety set

Listing 16.2.5.3 - Dose per body weight - Safety set

Listing 16.2.5.4 - PK samples collection dates and times

Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

Listing 16.2.7.1 - Treatment-emergent adverse events

Listing 16.2.7.2 - Pre-treatment adverse events

Listing 16.2.8.1 - Individual laboratory measurements

Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

Listing 16.2.9.1 - Vital signs and body weight

Listing 16.2.9.2 - Recorded parameters of ECG

Listing 16.2.9.3 - Investigator's interpretation of ECG

Listing 16.2.10.1 - Medical and surgical history

Listing 16.2.10.2 - Physical examination

Sponsor code PNET-22-08 Netupitant IV infusion shortening Final version 1.0, 18JUN24

Statistical analysis plan CRO-PK-22-363




# CROSS ALLIANCE Contract Research Organisation for Scientific Services

## Section 16.2 - Individual Subject Data Listings Shells

Listing 16.2.10.3 - Prior and concomitant medications

Listing 16.2.10.4 - Substance use

Listing 16.2.10.5 - Subjects study visits

Listing 16.2.10.6 - Fertility status and contraception

Listing 16.2.10.7 - Reproductive status and contraception

Listing 16.2.10.8 - Meals



# **Listing 16.2.1.1 - Discontinued subjects**

| Subject<br>ID | Cohort | Sex | Age<br>(years) | Last<br>visit | Date/time of<br>last IMP<br>administration | Date of premature Study termination | Time elapsed from<br>last IMP<br>administration<br>(days) | Primary reason for subject premature study termination |
|---|---|---|---|---|---|---|---|---|
| S001/001 | 1: 30 min (Rα) | F | 22 | Visit 3 - Days 1-2 | ddMMMyyyy hh:mm | ddMMMyyyy | 1 | Withdrawal by subject |
| S012/011 | 2: 30 min (T) | M | 40 | Visit 3 - Days 1-2 | ddMMMyyyy hh:mm | ddMMMyyyy | 1 | Adverse event |
| | | | | | ••• | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



**Listing 16.2.2.1 - Protocol deviations** 

| Subject<br>ID | Cohort | Deviation<br>Number | Deviation<br>Category | Deviation<br>Coded<br>Term | Deviation<br>Description |
|---|---|---|---|---|---|
| S001/001 | 1: 30 min (Rα) | 1 | Minor | Deviation from scheduled sampling time | Sample number 2 was collected outside the window of 30 min pre-dose |
| S019/016 | 1: 30 min (T) | 1 | Major | Inclusion criteria violation | Inclusion criteria violation |
| S026/022 | 2: 15 min (T) | 1 | Major | Inclusion criteria violation | Inclusion criteria violation |
| S039/033 | 3: 5 min (T) | 1 | Minor | Deviation in EGC recording | Deviation occurred during collection of EGC recording |
| S047/041 | 4: 2 min (T) | 1 | Minor | Deviation from scheduled sampling time | Sample number 2 was collected outside the window of 30 min pre-dose |
| | ••• | | | | |

Program: Listings\k363-dv-lst.sas


Listing 16.2.3.1 - Subjects excluded from safety and/or PK analysis

| Subject<br>ID | Cohort | Sex | Age<br>(vears) | Enrolled<br>Set | Safety<br>Set | PK<br>Set | Reason for the exclusion |
|---|---|---|---|---|---|---|---|
| | 1 20 · (T) | | | | ) I | N. | I 1 CD (D' + 1 (C C + 1) N DV 1 + 111 (DV +) |
| S14/012 | 1: 30 min (T) | F | 23 | Y | N | N | Lack of IMP intake (Safety set); No PK data available (PK set) |
| S37/032 | 3: 5 min (T) | F | 52 | Y | Y | N | No PK data available (PK set) |
| | ••• | ••• | | ••• | ••• | ••• | |

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Enrolment | Date of<br>Administration | Completed<br>or<br>Discontinued | Date of<br>End of Study | Reason for discontinuation |
|---|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | Withdrawal by subject |
| ••• | | ••• | | ••• | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

**Cohort 1: 30 min (T)** 

| | Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Enrolment | Date of<br>Administration | Completed<br>or<br>Discontinued | Date of<br>End of Study | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| _ | S013/011 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | |
| | ••• | ••• | ••• | ••• | ••• | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

**Cohort 2: 15 min (T)** 

| | Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Enrolment | Date of<br>Administration | Completed<br>or<br>Discontinued | Date of<br>End of Study | Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| _ | S024/021 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | Adverse event |
| | | ••• | ••• | ••• | ••• | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

Cohort 3: 5 min (T)

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Enrolment | Date of<br>Administration | Completed<br>or<br>Discontinued | Date of<br>End of Study | Reason for discontinuation |
|---|---|---|---|---|---|---|---|
| S038/031 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | Withdrawal by subject |
| | | ••• | | ••• | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

Cohort 4: 2 min (T)

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Enrolment | Date of<br>Administration | Completed<br>or<br>Discontinued | Date of<br>End of Study | Reason for discontinuation |
|---|---|---|---|---|---|---|---|
| S049/041 | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ds-lst.sas



# Listing 16.2.4.2 - Demography

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Sex | Birth<br>Year | Ethnicity | Race | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| S001/001 | F | 1983 | Not Hispanic or Latino | White | 40 | 170 | 55.0 | 18.0 |
| | | | ••• | ••• | | | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to \_

Program:Listings\k363-dm-lst.sas



# **Listing 16.2.4.2 - Demography**

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Sex | Birth<br>Year | Ethnicity | Race | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| S002/002 | F | 1990 | Hispanic or Latino | Other | 33 | 165 | 65.0 | 23.9 |
| ••• | ••• | ••• | ••• | ••• | | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to \_

Program:Listings\k363-dm-lst.sas



# Listing 16.2.4.2 - Demography

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Sex | Birth<br>Year | Ethnicity | Race | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| S024/021 | M | 1978 | Not Hispanic or Latino | White | 45 | 180 | 85.0 | 26.2 |
| | ••• | ••• | ••• | ••• | | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to \_

Program:Listings\k363-dm-lst.sas



# Listing 16.2.4.2 - Demography

# Cohort 3: 5 min (T)

| Subject<br>ID | Sex | Birth<br>Year | Ethnicity | Race | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| S035/031 | M | 1992 | Not Hispanic or Latino | White | 29 | 177 | 75.0 | 23.9 |
| ••• | ••• | ••• | ••• | ••• | | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to \_

Program:Listings\k363-dm-lst.sas



# Listing 16.2.4.2 - Demography

# Cohort 4: 2 min (T)

| Subject<br>ID | Sex | Birth<br>Year | Ethnicity | Race | Age<br>(years) | Height (cm) | Body Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| S048/041 | F | 1975 | Not Hispanic or Latino | White | 48 | 163 | 59.0 | 22.2 |
| ••• | ••• | | ••• | ••• | | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to \_

Program:Listings\k363-dm-lst.sas



Listing 16.2.4.3 - Inclusion/Exclusion criteria not met

| Subject<br>ID | Cohort | Criterion | Verbatim |
|---|---|---|---|
| S001/001 | 1: 30 min (Rα) | Exclusion criterion 3 | Laboratory analyses: laboratory values clinically significant abnormal at screening, indicative of physical illness or suggesting the subject's exclusion, in his/her best interest |
| 015/012 | 1: 30 min (T) | Exclusion criterion 9 | Blood donation or significant blood loss: blood donations or significant blood loss in the 3 months before the first visit of this study |
| 028/023 | 2: 15 min (T) | Exclusion criterion 14 | Positive or missing pregnancy test at screening or Day -1, pregnant or lactating women |
| 037/032 | 3: 5 min (T) | Exclusion criterion 3 | Clinically significant abnormal laboratory values at screening, indicative of physical illness or suggesting the subject's exclusion, in his/her best interest |
| 049/043 | 4: 2 min (T) | Exclusion criterion 2 | Clinically significant abnormal physical findings which could interfere with the objectives of the study |
| | ••• | | |

Program: Listings\k363-ie-lst.sas



# Listing 16.2.4.4 - Physical examination at screening

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | Body System | Interpretation | Findings |
|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | General Appearance | Normal | |
| | | | Head, Eyes, Ears, Nose and Throat | Normal | |
| | | | Skin | Abnormal, not Clinical significant | Left wrist cicatrix |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pe-lst.sas



# Listing 16.2.4.4 - Physical examination at screening

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | Body System | Interpretation | Findings |
|---|---|---|---|---|---|
| S013/011 | Screening | ddMMMyyyy | General Appearance | Normal | |
| | | | Head, Eyes, Ears, Nose and Throat | Normal | |
| | ••• | ••• | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pe-lst.sas



# Listing 16.2.4.4 - Physical examination at screening

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | Body System | Interpretation | Findings |
|---|---|---|---|---|---|
| S24/021 | Screening | ddMMMyyyy | General Appearance | Normal | |
| | | | Head, Eyes, Ears, Nose and Throat | Normal | |
| | | ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pe-lst.sas



# Listing 16.2.4.4 - Physical examination at screening

Cohort 3: 5 min (T)

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | Body System | Interpretation | Findings |
|---|---|---|---|---|---|
| S35/031 | Screening | ddMMMyyyy | General Appearance | Normal | |
| | | | Head, Eyes, Ears, Nose and Throat | Normal | |
| ••• | ••• | ••• | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pe-lst.sas



# Listing 16.2.4.4 - Physical examination at screening

Cohort 4: 2 min (T)

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | Body System | Interpretation | Findings |
|---|---|---|---|---|---|
| S46/041 | Screening | ddMMMyyyy | General Appearance | Normal | |
| | | | Head, Eyes, Ears, Nose and Throat | Normal | |
| ••• | ••• | ••• | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pe-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time Point | Date/Time of<br>Start of<br>Administration | Date/Time of<br>End of<br>Administration | Volume<br>Administered<br>(mL) | Has there been at least one interruption? | Interruption<br>Nr. | Was the interruption due to AE? | Time of Start of<br>Interruption | Time of End of<br>Interruption |
|---|---|---|---|---|---|---|---|---|---|
| S001/001 | Visit 3 | ddMMMyyyy<br>hh:mm | ddMMMyyyy<br>hh:mm | 20 | Y | 1 | N | hh:mm | hh:mm |
| ••• | | ••• | ••• | ••• | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time Point | Date/Time of<br>Start of<br>Administration | Date/Time of<br>End of<br>Administration | Volume<br>Administered<br>(mL) | Has there been at least one interruption? | Interruption<br>Nr. | Was the interruption due to AE? | Time of Start of<br>Interruption | Time of End of<br>Interruption |
|---|---|---|---|---|---|---|---|---|---|
| S012/011 | Visit 3 | ddMMMyyyy<br>hh:mm | ddMMMyyyy<br>hh:mm | 20 | Y | 1 | N | hh:mm | hh:mm |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time Point | Date/Time of<br>Start of<br>Administration | Date/Time of<br>End of<br>Administration | Volume<br>Administered<br>(mL) | Has there been at least one interruption? | Interruption<br>Nr. | Was the interruption due to AE? | Time of Start of<br>Interruption | Time of End of<br>Interruption |
|---|---|---|---|---|---|---|---|---|---|
| S024/021 | Visit 3 | ddMMMyyyy<br>hh:mm | ddMMMyyyy<br>hh:mm | 20 | N | NA | NA | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

Cohort 3: 5 min (T)

| Subject<br>ID | Time Point | Date/Time of<br>Start of<br>Administration | Date/Time of<br>End of<br>Administration | Volume<br>Administered<br>(mL) | Has there been at least one interruption? | Interruption<br>Nr. | Was the interruption due to AE? | Time of Start of<br>Interruption | Time of End of<br>Interruption |
|---|---|---|---|---|---|---|---|---|---|
| S035/031 | Visit 3 | ddMMMyyyy<br>hh:mm | ddMMMyyyy<br>hh:mm | 20 | N | NA | NA | | |
| | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.1 - Investigational medicinal products administration

Cohort 4: 2 min (T)

| Subject<br>ID | Time Point | Date/Time of<br>Start of<br>Administration | Date/Time of<br>End of<br>Administration | Volume<br>Administered<br>(mL) | Has there been at least one interruption? | Interruption<br>Nr. | Was the interruption due to AE? | Time of Start of<br>Interruption | Time of End of<br>Interruption |
|---|---|---|---|---|---|---|---|---|---|
| S046/041 | Visit 3 | ddMMMyyyy<br>hh:mm | ddMMMyyyy<br>hh:mm | 20 | N | NA | NA | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# **Listing 16.2.5.2 - Fasting conditions**

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time Point | Date/Time of<br>Start of Administration | Fasting Conditions From 10 h before IMP Administration? | Fasting Conditions<br>Start Date/time | Duration between Start of Fasting Conditions and Start of IMP administration |
|---|---|---|---|---|---|
| S001/001 | Visit 3 | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm | xx h xx min |
| ••• | ••• | ··· | ··· | ··· | ···· |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# **Listing 16.2.5.2 - Fasting conditions**

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time Point | Date/Time of<br>Start of Administration | Fasting Conditions<br>From 10 h before<br>IMP Administration? | Fasting Conditions<br>Start Date/time | Duration between Start of Fasting Conditions and Start of IMP administration |
|---|---|---|---|---|---|
| S012/011 | Visit 3 | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm | xx h xx min |
| ••• | ••• | | | ··· | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# **Listing 16.2.5.2 - Fasting conditions**

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time Point | Date/Time of<br>Start of Administration | Fasting Conditions From 10 h before IMP Administration? | Fasting Conditions<br>Start Date/time | Duration between Start of Fasting Conditions and Start of IMP administration |
|---|---|---|---|---|---|
| S024/021 | Visit 3 | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm | xx h xx min |
| ••• | ••• | | ··· | ··· | ···· |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# **Listing 16.2.5.2 - Fasting conditions**

Cohort 3: 5 min (T)

| Subject<br>ID | Time Point | Date/Time of<br>Start of Administration | Fasting Conditions From 10 h before IMP Administration? | Fasting Conditions<br>Start Date/time | Duration between Start of Fasting Conditions and Start of IMP administration |
|---|---|---|---|---|---|
| S035/031 | Visit 3 | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm | xx h xx min |
| ••• | ••• | | | ··· | ···· |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# **Listing 16.2.5.2 - Fasting conditions**

Cohort 4: 2 min (T)

| Subject<br>ID | Time Point | Date/Time of<br>Start of Administration | Fasting Conditions From 10 h before IMP Administration? | Fasting Conditions<br>Start Date/time | Duration between Start of Fasting Conditions and Start of IMP administration |
|---|---|---|---|---|---|
| S046/041 | Visit 3 | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm | xx h xx min |
| ••• | ••• | | ··· | ··· | ···· |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.3 - Dose per body weight

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Active Ingredient | Dose per<br>Administration<br>(mg) | Body Weight (kg) | Dose per<br>Body Weight<br>(mg/kg) |
|---|---|---|---|---|
| S001/001 | Fosnetupitant | 235 | 55.0 | 4.27 |
| S001/001 | Palonosetron | 0.25 | 55.0 | 0.005 |

Note: Subjects are listed according to the cohort they belong to

The dose per body weight is calculated using the screening body weight and the actual dose administered

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.3 - Dose per body weight

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Active Ingredient | Dose per<br>Administration<br>(mg) | Body Weight (kg) | Dose per<br>Body Weight<br>(mg/kg) |
|---|---|---|---|---|
| S012/011 | Fosnetupitant | 235 | 70.0 | 3.36 |
| ••• | ••• | ··· | ···· | ···· |

Note: Subjects are listed according to the cohort they belong to

The dose per body weight is calculated using the screening body weight and the actual dose administered

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.3 - Dose per body weight

**Cohort 1: 15 min (T)** 

| Subject<br>ID | <b>Active Ingredient</b> | Dose per<br>Administration | Body Weight (kg) | Dose per<br>Body Weight |
|---|---|---|---|---|
| | | (mg) | (8) | (mg/kg) |
| S024/021 | Fosnetupitant | 235 | 70.0 | 3.36 |

Note: Subjects are listed according to the cohort they belong to

The dose per body weight is calculated using the screening body weight and the actual dose administered

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.3 - Dose per body weight

Cohort 1: 5 min (T)

| Subject<br>ID | Active Ingredient | Dose per<br>Administration<br>(mg) | Body Weight (kg) | Dose per<br>Body Weight<br>(mg/kg) |
|---|---|---|---|---|
| S036/031 | Fosnetupitant | 235 | 64.0 | 3.67 |
| ••• | ••• | | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

The dose per body weight is calculated using the screening body weight and the actual dose administered

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.3 - Dose per body weight

Cohort 1: 2 min (T)

| Subject<br>ID | Active Ingredient | Dose per<br>Administration<br>(mg) | Body Weight (kg) | Dose per<br>Body Weight<br>(mg/kg) |
|---|---|---|---|---|
| S048/041 | Fosnetupitant | 235 | 57.0 | 4.12 |
| ••• | <b></b> | <b></b> | <b></b> | ···· |

Note: Subjects are listed according to the cohort they belong to

The dose per body weight is calculated using the screening body weight and the actual dose administered

Program: Listings\k363-ex-lst.sas



# Listing 16.2.5.4 - PK samples collection dates and times

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | IMP<br>Administration | Sample<br>Number | Nominal<br>Time Point | Collection Date/time | Time from the start of IMP | Sampling collection time as |
|---|---|---|---|---|---|---|
| | Start Date/Time | | | | infusion/injection | per protocol? |
| S001/001 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before start of infusion | ddMMMyyyy hh:mm | -xx min | Yes |
| S001/001 | ddMMMyyyy hh:mm | 2 | 30 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S001/001 | ddMMMyyyy hh:mm | 3 | 45 min $\pm$ 2 min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| S001/001 | ddMMMyyyy hh:mm | 4 | 1 h $\pm$ 2 min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| S001/001 | ddMMMyyyy hh:mm | 5 | $1.5h \pm 2$ min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| | ••• | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pc-lst.sas



# Listing 16.2.5.4 - PK samples collection dates and times

**Cohort 1: 30 min (T)** 

| Subject<br>ID | IMP<br>Administration<br>Start Date/Time | Sample<br>Number | Nominal<br>Time Point | Collection<br>Date/time | Time from<br>the start of IMP<br>infusion/injection | Sampling collection<br>time as<br>per protocol? |
|---|---|---|---|---|---|---|
| S012/011 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before start of infusion | ddMMMyyyy hh:mm | -xx min | Yes |
| S012/011 | ddMMMyyyy hh:mm | 2 | 30 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S012/011 | ddMMMyyyy hh:mm | 3 | $45 \min \pm 2 \min$ after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| S012/011 | ddMMMyyyy hh:mm | 4 | 1 h $\pm$ 2 min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| S012/011 | ddMMMyyyy hh:mm | 5 | $1.5h \pm 2$ min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| | ••• | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pc-lst.sas



# Listing 16.2.5.4 - PK samples collection dates and times

**Cohort 2: 15 min (T)** 

| Subject<br>ID | IMP<br>Administration | Sample<br>Number | Nominal<br>Time Point | Collection Date/time | Time from the start of IMP | Sampling collection time as |
|---|---|---|---|---|---|---|
| | Start Date/Time | | | | infusion/injection | per protocol? |
| S024/021 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before start of infusion | ddMMMyyyy hh:mm | -xx min | Yes |
| S024/021 | ddMMMyyyy hh:mm | 2 | 15 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S024/021 | ddMMMyyyy hh:mm | 3 | 20 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S024/021 | ddMMMyyyy hh:mm | 4 | 30 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S024/021 | ddMMMyyyy hh:mm | 5 | 45 min $\pm$ 2 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| | ••• | | | | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pc-lst.sas



# Listing 16.2.5.4 - PK samples collection dates and times

# Cohort 3: 5 min (T)

| Subject<br>ID | IMP<br>Administration<br>Start Date/Time | Sample<br>Number | Nominal<br>Time Point | Collection<br>Date/time | Time from<br>the start of IMP<br>infusion/injection | Sampling collection time as per protocol? |
|---|---|---|---|---|---|---|
| S036/031 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before start of infusion | ddMMMyyyy hh:mm | -xx min | No |
| S036/031 | ddMMMyyyy hh:mm | 2 | 5 min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| S036/031 | ddMMMyyyy hh:mm | 3 | 10 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S036/031 | ddMMMyyyy hh:mm | 4 | 15 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S036/031 | ddMMMyyyy hh:mm | 5 | 20 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| | | ••• | <b></b> | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pc-lst.sas


# Listing 16.2.5.4 - PK samples collection dates and times

# Cohort 4: 2 min (T)

| Subject<br>ID | IMP<br>Administration<br>Start Date/Time | Sample<br>Number | Nominal<br>Time Point | Collection<br>Date/time | Time from<br>the start of IMP<br>infusion/injection | Sampling collection<br>time as<br>per protocol? |
|---|---|---|---|---|---|---|
| S048/041 | ddMMMyyyy hh:mm | 1 | Pre-dose - Within 30 min before start of infusion | ddMMMyyyy hh:mm | -xx min | Yes |
| S048/041 | ddMMMyyyy hh:mm | 2 | 2 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S048/041 | ddMMMyyyy hh:mm | 3 | 5 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S048/041 | ddMMMyyyy hh:mm | 4 | 10 min after start of infusion | ddMMMyyyy hh:mm | xx min | Yes |
| S048/041 | ddMMMyyyy hh:mm | 5 | 15 min after start of infusion | ddMMMyyyy hh:mm | xx min | No |
| | ••• | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

#### **Cohort 1: 30 min (Rα)**

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | | | | | | | | ••• | | | ••• | ••• | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

**Cohort 1: 30 min (T)** 

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <br>S012/011 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | ••• | ••• | | ••• | ••• | ••• | ••• | | ••• | | | | ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

# **Cohort 2: 15 min (T)**

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

# Cohort 3: 5 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | ••• | ••• | | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.5 - Fosnetupitant Concentrations (ng/mL) measured in plasma

# Cohort 4: 2 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

#### **Cohort 1: 30 min (Rα)**

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | | | | | | | | ••• | | | ••• | ••• | | | ••• |

Note: Subjects are listed according to the cohort they belong to Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

# **Cohort 2: 15 min (T)**

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

# Cohort 3: 5 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | ••• | | | | ••• | ••• | | | ••• | ••• | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.6 - Netupitant Concentrations (ng/mL) measured in plasma

# Cohort 4: 2 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

#### **Cohort 1: 30 min (Rα)**

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <br>S001/001 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

# **Cohort 2: 15 min (T)**

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

# Cohort 3: 5 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.7 - Netupitant metabolite M1 Concentrations (ng/mL) measured in plasma

# Cohort 4: 2 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | | ••• | ••• | | | | | | ••• | | | | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

#### **Cohort 1: 30 min (Rα)**

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <br>S001/001 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

**Cohort 1: 30 min (T)** 

| | bject<br>D | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S01 | 2/011 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | ••• | | | ••• | ••• | | | ••• | ••• | | ••• | ••• | | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | ••• | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | | | ••• | ••• | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

# Cohort 3: 5 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.8 - Netupitant metabolite M2 Concentrations (ng/mL) measured in plasma

# Cohort 4: 2 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | | | ••• | ••• | | | | | | ••• | | | | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

#### **Cohort 1: 30 min (Rα)**

| <br>Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <br>S001/001 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | ••• | ••• | ••• | ••• | ••• | ••• | | ••• | ••• | | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

**Cohort 1: 30 min (T)** 

| | bject<br>D | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S01 | 2/011 | XX.XX | | | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | ••• | | | ••• | ••• | | | ••• | ••• | | ••• | ••• | | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

# **Cohort 2: 15 min (T)**

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XX.XX | | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| ••• | | ••• | | ••• | | | | | ••• | | | | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



#### Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

# Cohort 3: 5 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XX.XX | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



### Listing 16.2.5.9 - Netupitant metabolite M3 Concentrations (ng/mL) measured in plasma

# Cohort 4: 2 min (T)

| Subject<br>ID | Pre<br>dose | 2 min | 5 min | 10 min | 15 min | 20 min | 30 min | 45 min | 1 hour | 1.5 hour | 2 h | 3 h | 4 h | 8 h | 12 h | 24 h |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | | | | ••• | ••• | ••• | ••• | | ••• | | ••• | | ••• | | ••• |

Note: Subjects are listed according to the cohort they belong to

Sampling times are counted from the start of the injection/infusion

BQL: Below Lower Quantification Limit (20.00 ng/mL)

Program: Listings\k363-pc-lst.sas



# Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub><br>(ng/mL) | tı <sub>ast</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

**Cohort 1: 30 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | ••• | | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

**Cohort 2: 15 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| ••• | | | | | ••• | | | ••• | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Cohort 3: 5 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.1 - Plasma PK parameters - Fosnetupitant

Cohort 4: 2 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | ••• | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.2 - Plasma PK parameters - Netupitant

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub><br>(ng/mL) | t <sub>last</sub> (h) | t <sub>max</sub><br>(h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| ••• | | | | | | | | ••• | | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.2 - Plasma PK parameters - Netupitant

**Cohort 1: 30 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\begin{array}{c} \lambda_z \\ (1/h) \end{array}$ | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | ••• | ••• | ••• | ••• | ••• | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.2 - Plasma PK parameters - Netupitant

**Cohort 2: 15 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| ••• | | | | | ••• | ••• | | ••• | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Cohort 3: 5 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.2 - Plasma PK parameters - Netupitant

Cohort 4: 2 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\begin{array}{c} \lambda_z \\ (1/h) \end{array}$ | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas


# Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

### **Cohort 1: 30 min (Rα)**

| Subject | $\mathbf{C}_{\max}$ | Co | Clast | tlast | tmax | <b>AUC</b> last | <b>AUC</b> 0-24 | $\lambda_z$ | <b>t</b> ½ | $\mathbf{CL}$ | $V_z$ | MRT |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | (ng/mL) | (ng/mL) | (ng/mL) | (h) | (h) | (h*ng/mL) | (h*ng/mL) | (1/h) | (h) | (mL/h) | (mL) | (h) |
| S001/001 | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX |
| | | | | | | ••• | | | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

**Cohort 1: 30 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub> (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx |
| ••• | | | | | ••• | | | ••• | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

**Cohort 2: 15 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | ••• | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

Cohort 3: 5 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.3 - Plasma PK parameters - Netupitant metabolite M1

Cohort 4: 2 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | ••• | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub><br>(ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

**Cohort 1: 30 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | ••• | | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

**Cohort 2: 15 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | ••• | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

Cohort 3: 5 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.4 - Plasma PK parameters - Netupitant metabolite M2

Cohort 4: 2 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | ••• | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | C <sub>last</sub><br>(ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub><br>(h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S001/001 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

**Cohort 1: 30 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\begin{array}{c} \lambda_z \\ (1/h) \end{array}$ | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S012/011 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | ••• | ••• | | ••• | ••• | | | ••• | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

**Cohort 2: 15 min (T)** 

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT<br>(h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S024/021 | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xxx.xx | XXX.XX | xxx.xx |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

Cohort 3: 5 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | Vz<br>(mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S036/031 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



# Listing 16.2.6.5 - Plasma PK parameters - Netupitant metabolite M3

Cohort 4: 2 min (T)

| Subject<br>ID | C <sub>max</sub> (ng/mL) | C <sub>0</sub> (ng/mL) | Clast (ng/mL) | t <sub>last</sub><br>(h) | t <sub>max</sub> (h) | AUC <sub>last</sub> (h*ng/mL) | AUC <sub>0-24</sub> (h*ng/mL) | $\lambda_z$ (1/h) | t½<br>(h) | CL<br>(mL/h) | $V_z$ (mL) | MRT (h) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| S048/041 | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | ••• | | | | | | | ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: pk-analysis\k363-pp-lst.sas



### Listing 16.2.7.1 - Treatment-emergent adverse events

### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Adverse<br>Event | | |
|---|---|---|---|
| | ID | | |
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class 1: | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



### Listing 16.2.7.1 - Treatment-emergent adverse events

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S012/011 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



### Listing 16.2.7.1 - Treatment-emergent adverse events

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S024/021 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | <del></del> |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| | | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



### Listing 16.2.7.1 - Treatment-emergent adverse events

Cohort 3: 5 min (T)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S036/031 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



### Listing 16.2.7.1 - Treatment-emergent adverse events

Cohort 4: 2 min (T)

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S048/041 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Last Study Drug Administration Date/Time Before Onset: | ddMMMyyyy hh:mm |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | None |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

### **Cohort 1: 30 min (Rα)**

| Subject | | | |
|---|---|---|---|
| ID | Event<br>ID | | |
| S001/001 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S012/011 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | <del></del> |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Adverse<br>Event<br>ID | | |
|---|---|---|---|
| S024/021 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

Cohort 3: 5 min (T)

| Subject<br>ID | Adverse<br>Event | | |
|---|---|---|---|
| 12 | ID | | |
| S036/031 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |
| ••• | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

Cohort 4: 2 min (T)

| Subject<br>ID | Adverse<br>Event | | |
|---|---|---|---|
| ID | ID | | |
| S048/041 | 1 | Description: | Headache |
| | | Preferred Term <sup>1</sup> : | Headache |
| | | System Organ Class <sup>1</sup> : | Nervous system disorders |
| | | Start Date/Time - End Date/Time (Day): | ddMMMyyyy hh:mm (k) - ddMMMyyyy (j) |
| | | Relation to the Study Drug | Not related |
| | | Severity: | Mild |
| | | Serious Adverse Event? | N |
| | | Seriousness criteria: | |
| | | Action Taken with Study Drug: | |
| | | Other Action Taken: | None |
| | | Outcome: | Recovered/Resolved |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-ae-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |
| ••• | ••• | | | ••• | ••• | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |

Note: Subjects are listed according to the cohort they belong to

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | | ••• | | ••• |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | ••• | <b></b> | | ••• | ••• |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: URINE DRUG SCREENING** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S001/001 | Screening | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| ••• | ••• | ••• | | ••• | ••• | ••• |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative | Negative | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative | Negative | NCS |
| S001/001 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative | Negative | NCS |
| ••• | | | <b></b> | | ••• | |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (Rα)** 

Category of Laboratory Parameters: SALIVARY BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Pregnancy Test (Serum) | Negative | Negative | NCS |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test (Urine) | Negative | Negative | |
| S001/001 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Salivary Alcohol Test | Negative | Negative | |
| ••• | ••• | ••• | <b></b> | ••• | ••• | |

Note 1: A=Different from reference value

Note 2: Clinical Significance is reported for serum pregnancy test only. CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |
| | | | | ••• | ••• | ••• |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | <b></b> | | | |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10 <sup>12</sup> /L] | 5.19 | 3.90 - 5.30 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | | | | ••• | |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | | | | | ••• |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: URINE DRUG SCREENING** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S012/011 | Screening | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| ••• | | | <b></b> | ••• | ••• | ••• |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative | Negative | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative | Negative | NCS |
| S012/011 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative | Negative | NCS |
| | | | <b></b> | ••• | ••• | |

Note 1: A=Different from reference value

Note 2: Clinical Significance is reported for serum pregnancy test only. CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas


### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 1: 30 min (T)** 

Category of Laboratory Parameters: SALIVARY BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Pregnancy Test (Serum) | Negative | Negative | NCS |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test (Urine) | Negative | Negative | |
| S012/011 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Salivary Alcohol Test | Negative | Negative | |
| ••• | | ••• | ··· | ••• | | ••• |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |
| ••• | | ••• | | ••• | ••• | |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10 <sup>12</sup> /L] | 5.19 | 3.90 - 5.30 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | <b></b> | | | |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | | | ••• | |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | | <b></b> | | ••• | |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | | | ••• | | |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: URINE DRUG SCREENING** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S024/021 | Screening | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| ••• | | | | ••• | ••• | |

Note 1: A=Different from reference value

Note 2: Clinical Significance is reported for serum pregnancy test only. CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative | Negative | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative | Negative | NCS |
| S024/021 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative | Negative | NCS |
| ••• | ••• | ••• | <b></b> | | ••• | ••• |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

**Cohort 2: 15 min (T)** 

Category of Laboratory Parameters: SALIVARY BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Pregnancy Test (Serum) | Negative | Negative | NCS |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test (Urine) | Negative | Negative | |
| S024/021 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Salivary Alcohol Test | Negative | Negative | |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |
| | | | | ••• | | ••• |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10 <sup>12</sup> /L] | 5.19 | 3.90 - 5.30 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | <b></b> | | | |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | ••• | <b></b> | | | |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| | | ••• | | | | |

Note 1: A=Different from reference value

Note 2: Clinical Significance is reported for serum pregnancy test only. CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: URINE DRUG SCREENING** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S036/031 | Screening | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| | | | | ••• | | |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



#### **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 3: 5 min (T)

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative | Negative | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative | Negative | NCS |
| S036/031 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative | Negative | NCS |
| ••• | ••• | <b></b> | | ••• | ••• | ••• |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

## Cohort 3: 5 min (T)

Category of Laboratory Parameters: SALIVARY BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Pregnancy Test (Serum) | Negative | Negative | NCS |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test (Urine) | Negative | Negative | |
| S036/031 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Salivary Alcohol Test | Negative | Negative | |
| ••• | | ••• | <b></b> | ••• | | ••• |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: BLOOD CHEMISTRY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |
| | | | | ••• | | ••• |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Sodium [mmol/L] | 138 | 136 - 145 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Potassium [mmol/L] | 4.4 | 3.5 - 5.1 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Calcium [mmol/L] | 2.27 | 2.10 - 2.55 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Chloride [mmol/L] | 103 | 96 - 110 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Phosphate [mmol/L] | 0.84 [A] | 0.87 - 1.45 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Alkaline Phosphatase [U/L] | 95 | <= 104 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Gamma Glutamyl Transferase [U/L] | 17 | <= 39 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Aspartate Aminotransferase [U/L] | 24 | <= 35 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Alanine Aminotransferase [U/L] | 30 | <= 35 | NCS |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: HAEMATOLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | | | *** | |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Leukocytes [10^9/L] | 10.02 [A] | 4.00 - 10.00 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Erythrocytes [10^12/L] | 5.19 | 3.90 - 5.30 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [g/dL] | 15.4 | 12.0 - 16.0 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Hemoglobin [mmol/L] | 9.6 | 7.5 - 9.9 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Hematocrit [%] | 44 | 37 - 47 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Volume [fL] | 84 | 83 - 100 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular Hemoglobin [pg] | 30 | 27 - 34 | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Ery. Mean Corpuscular HGB Concentration [g/dL] | 35 | 32 - 36 | NCS |
| | | | | | | ••• |

Note 1: A=Different from reference value

Note 2: Clinical Significance is reported for serum pregnancy test only. CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: URINE ANALYSIS** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urobilinogen | Normal | Normal | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urinary Bilirubin | Absent | Absent | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Ketones | Absent | Absent | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urinary Hemoglobin | +++ [A] | Absent | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urinary Leukocytes | Absent | Absent | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Sediment Examination | Checked | | |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Leukocytes | Absent | Absent or 0-2 per field | NCS |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Urinary Sediment Erythrocytes | 0-2 per field | Absent or 0-2 per field | NCS |

Note 1: A=Abnormal

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



## **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: URINE DRUG SCREENING** 

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S048/041 | Screening | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Amphetamine | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cannabinoids | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Cocaine | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Ecstasy | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Methamphetamine | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Opiate | Negative | Negative | |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

Cohort 4: 2 min (T)

**Category of Laboratory Parameters: VIROLOGY** 

| Subject<br>ID | Time<br>Point | Collection<br>Date/time | Parameter | Value and Abnormality <sup>1</sup> | Normal Range or<br>Reference Value | Clinically<br>Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Hepatitis B Virus Surface Antigen | Negative | Negative | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | Hepatitis C Virus Antibody | Negative | Negative | NCS |
| S048/041 | Screening | ddMMMyyyy hh:mm | HIV Ag/Ab Combo | Negative | Negative | NCS |
| ••• | | | <b></b> | ••• | ••• | ••• |

Note 1: A=Different from reference value

Note 2: Clinical Significance is not collected for Urine Drug Screening

Program: Listings\k363-lb-lst.sas



### **Listing 16.2.8.1 - Individual laboratory measurements**

## Cohort 4: 2 min (T)

Category of Laboratory Parameters: SALIVARY BREATH TEST AND PREGNANCY TEST

| Subject<br>ID | Time<br>Point | Collection Date/time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range or Reference Value | Clinically Significant? <sup>2</sup> |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Pregnancy Test (Serum) | Negative | Negative | NCS |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Pregnancy Test (Urine) | Negative | Negative | |
| S048/041 | Visit 2 - Day -1 | ddMMMyyyy hh:mm | Salivary Alcohol Test | Negative | Negative | |
| | | ••• | | ••• | ••• | ••• |

Note 1: A=Different from reference value

Note 2: CS= Clinically Significant, NCS= Not Clinically Significant

Program: Listings\k363-lb-lst.sas



# Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

## **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Assessment<br>Date | Specimen | Investigator's<br>Interpretation | Which AE the Abnormality is related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy | Blood | Abnormal, Not Clinically Significant | | |
| S001/001 | Screening | ddMMMyyyy | Urine | Abnormal, Not Clinically Significant | | <del></del> |
| S001/001 | End of Study | ddMMMyyyy | Blood | Normal | | <del></del> |
| S001/001 | End of Study | ddMMMyyyy | Urine | Normal | | <del></del> |

Note: Subjects are listed according to the cohort they belong to

Note: End of Study = final visit or early termination visit

Program: Listings\k363-lb-lst.sas



# Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

# **Cohort 1: 30 min (T)**

| Subject<br>ID | Time<br>Point | Assessment Date | Specimen | Investigator's<br>Interpretation | Which AE the Abnormality is related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy | Blood | Abnormal, Not Clinically Significant | | |
| S012/011 | Screening | ddMMMyyyy | Urine | Abnormal, Not Clinically Significant | | |
| S012/011 | End of Study | ddMMMyyyy | Blood | Normal | | |
| S012/011 | End of Study | ddMMMyyyy | Urine | Normal | | <del></del> |

Note: Subjects are listed according to the cohort they belong to Note: End of Study = final visit or early termination visit

Program: Listings\k363-lb-lst.sas



# Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

**Cohort 2: 15 min (T)** 

| Subje<br>ID | ct Time<br>Point | Assessment<br>Date | Specimen | Investigator's<br>Interpretation | Which AE the Abnormality is related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|
| S024/0 | 21 Screening | ddMMMyyyy | Blood | Abnormal, Not Clinically Significant | | |
| S024/0 | 21 Screening | ddMMMyyyy | Urine | Abnormal, Not Clinically Significant | | |
| S024/0 | 21 End of Study | ddMMMyyyy | Blood | Normal | | <del></del> |
| S024/0 | 21 End of Study | ddMMMyyyy | Urine | Normal | | |

Note: Subjects are listed according to the cohort they belong to Note: End of Study = final visit or early termination visit

Program: Listings\k363-lb-lst.sas



# Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

# Cohort 3: 5 min (T)

| | ıbject<br>ID | Time<br>Point | Assessment Date | Specimen | Investigator's<br>Interpretation | Which AE the Abnormality is related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|---|
| S03 | 36/031 | Screening | ddMMMyyyy | Blood | Abnormal, Not Clinically Significant | | |
| S03 | 36/031 | Screening | ddMMMyyyy | Urine | Abnormal, Not Clinically Significant | | |
| S03 | 36/031 | End of Study | ddMMMyyyy | Blood | Normal | | |
| S03 | 36/031 | End of Study | ddMMMyyyy | Urine | Normal | | <del></del> |

Note: Subjects are listed according to the cohort they belong to Note: End of Study = final visit or early termination visit

Program: Listings\k363-lb-lst.sas



# Listing 16.2.8.2 - Investigator's interpretation of laboratory test results

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Assessment<br>Date | Specimen | Investigator's<br>Interpretation | Which AE the Abnormality is related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy | Blood | Abnormal, Not Clinically Significant | | |
| S048/041 | Screening | ddMMMyyyy | Urine | Abnormal, Not Clinically Significant | | |
| S048/041 | End of Study | ddMMMyyyy | Blood | Normal | | |
| S048/041 | End of Study | ddMMMyyyy | Urine | Normal | | |

Note: Subjects are listed according to the cohort they belong to Note: End of Study = final visit or early termination visit

Program: Listings\k363-lb-lst.sas



# Listing 16.2.9.1 - Vital signs and body weight

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S001/001 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S001/001 | Screening | ddMMMyyyy hh:mm | Height [cm] | 166 | NA |
| S001/001 | Screening | ddMMMyyyy hh:mm | BMI [kg/m^2] | 20.1 | NA |
| S001/001 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 2 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 2 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 2 | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S001/001 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |

Note: Subjects are listed according to the cohort they belong to \_

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

 $Program: Listings \verb|\k363-vs-lst.sas|$ 



# Listing 16.2.9.1 - Vital signs and body weight

## **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S001/001 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |

Note: Subjects are listed according to the cohort they belong to \_

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S012/011 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S012/011 | Screening | ddMMMyyyy hh:mm | Height [cm] | 166 | NA |
| S012/011 | Screening | ddMMMyyyy hh:mm | BMI [kg/m^2] | 20.1 | NA |
| S012/011 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 2 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 2 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 2 | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S012/011 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S012/011 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S012/011 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S024/021 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S024/021 | Screening | ddMMMyyyy hh:mm | Height [cm] | 166 | NA |
| S024/021 | Screening | ddMMMyyyy hh:mm | BMI [kg/m^2] | 20.1 | NA |
| S024/021 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 2 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 2 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 2 | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S024/021 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S024/021 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S024/021 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| ••• | | | | | |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

# Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Assessment<br>Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S036/031 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S036/031 | Screening | ddMMMyyyy hh:mm | Height [cm] | 166 | NA |
| S036/031 | Screening | ddMMMyyyy hh:mm | BMI [kg/m^2] | 20.1 | NA |
| S036/031 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 2 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 2 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 2 | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S036/031 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

## Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S036/031 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S036/031 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S048/041 | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Screening | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Screening | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S048/041 | Screening | ddMMMyyyy hh:mm | Height [cm] | 166 | NA |
| S048/041 | Screening | ddMMMyyyy hh:mm | BMI [kg/m^2] | 20.1 | NA |
| S048/041 | Visit 2 | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 2 | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 2 | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 2 | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S048/041 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - Pre dose | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - at the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



## Listing 16.2.9.1 - Vital signs and body weight

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Assessment Date/Time | Parameter | Value and<br>Abnormality <sup>1</sup> | Normal Range |
|---|---|---|---|---|---|
| S048/041 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - 1 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - 2 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - 4 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | Visit 3 - 24 h after the end of injection | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Systolic Blood Pressure [mmHg] | 96 [L] | 100-139 |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Diastolic Blood Pressure [mmHg] | 58 | 50-89 |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Heart Rate [beats/min] | 88 | 50-90 |
| S048/041 | End of Study | ddMMMyyyy hh:mm | Weight [kg] | 55.5 | NA |

Note: Subjects are listed according to the cohort they belong to

End of Study = final visit or early termination visit

Note 1: H=Higher than upper normal limit, L=Lower than lower normal limit

Program: Listings\k363-vs-lst.sas



# Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001<br>S001/001 | Screening | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001<br>S001/001 | ě | | •••• | | |
| | Screening | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

 $Program: Listings \backslash k363\text{-}eg\text{-}lst.sas$ 



# Listing 16.2.9.2 - Recorded parameters of ECG

## **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| ~~~ | | | | | |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |

Note: Subjects are listed according to the cohort they belong to

 $Program: Listings \backslash k363\text{-}eg\text{-}lst.sas$


### Listing 16.2.9.2 - Recorded parameters of ECG

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| | | | | | ••• |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |

Note: Subjects are listed according to the cohort they belong to

 $Program: Listings \backslash k363\text{-}eg\text{-}lst.sas$ 



### Listing 16.2.9.2 - Recorded parameters of ECG

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 1: 30 min (T)** 

| Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|
| End of Study | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| End of Study | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| End of Study | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| End of Study | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| End of Study | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| | Point End of Study | Point End of Study 2nd End of Study 2nd End of Study 2nd End of Study 3rd | PointDate/TimeEnd of Study2ndddMMMyyyy hh:mmEnd of Study2ndddMMMyyyy hh:mmEnd of Study2ndddMMMyyyy hh:mmEnd of Study3rdddMMMyyyy hh:mm | PointDate/TimeEnd of Study2ndddMMMyyyy hh:mmQT Interval [msec]End of Study2ndddMMMyyyy hh:mmQTcB Interval [msec]End of Study2ndddMMMyyyy hh:mmQTcF Interval [msec]End of Study3rdddMMMyyyy hh:mmHeart Rate [beats/min]End of Study3rdddMMMyyyy hh:mmRR Interval [msec]End of Study3rdddMMMyyyy hh:mmPR Interval [msec]End of Study3rdddMMMyyyy hh:mmQRS Duration [msec]End of Study3rdddMMMyyyy hh:mmQT Interval [msec]End of Study3rdddMMMyyyy hh:mmQT Interval [msec]End of Study3rdddMMMyyyy hh:mmQTcB Interval [msec] |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# **Cohort 2: 15 min (T)**

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

**Cohort 2: 15 min (T)** 

| Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|
| End of Study | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| End of Study | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| End of Study | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| End of Study | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| End of Study | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| End of Study | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| | Point End of Study | Point End of Study 2nd End of Study 2nd End of Study 2nd End of Study 3rd | PointDate/TimeEnd of Study2ndddMMMyyyy hh:mmEnd of Study2ndddMMMyyyy hh:mmEnd of Study2ndddMMMyyyy hh:mmEnd of Study3rdddMMMyyyy hh:mm | PointDate/TimeEnd of Study2ndddMMMyyyy hh:mmQT Interval [msec]End of Study2ndddMMMyyyy hh:mmQTcB Interval [msec]End of Study2ndddMMMyyyy hh:mmQTcF Interval [msec]End of Study3rdddMMMyyyy hh:mmHeart Rate [beats/min]End of Study3rdddMMMyyyy hh:mmRR Interval [msec]End of Study3rdddMMMyyyy hh:mmPR Interval [msec]End of Study3rdddMMMyyyy hh:mmQRS Duration [msec]End of Study3rdddMMMyyyy hh:mmQT Interval [msec]End of Study3rdddMMMyyyy hh:mmQT Interval [msec]End of Study3rdddMMMyyyy hh:mmQTcB Interval [msec] |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

### Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

### Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

### Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| | | ••• | ••• | <del></del> | |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | Heart Rate [beats/min] | xxx |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 1st | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.2 - Recorded parameters of ECG

# Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Parameter | Value |
|---|---|---|---|---|---|
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QT Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 2nd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | Heart Rate [beats/min] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | RR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | PR Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QRS Duration [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QT Interval [msec] | xxx |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcB Interval [msec] | XXX |
| S001/001 | End of Study | 3rd | ddMMMyyyy hh:mm | QTcF Interval [msec] | xxx |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.3 - Investigator's interpretation of ECG

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Investigator's<br>Interpretation | Investigator's<br>Comment | Which AE the<br>Abnormality is<br>related to? | Which MH the<br>Abnormality is<br>related to? |
|---|---|---|---|---|---|---|---|
| S001/001 | Screening | 1st | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S001/001<br>S001/001 | Screening | 2nd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S001/001<br>S001/001 | Screening | 3rd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| G004/004 | | | | | | | |
| S001/001 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S001/001 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S001/001 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Normal | | | |
| S001/001 | End of study | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S001/001 | End of study | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S001/001 | End of study | 3rd | ddMMMyyyy hh:mm | Normal | | | |

Note: Subjects are listed according to the cohort they belong to

NCS: Not Clinically Significant Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.3 - Investigator's interpretation of ECG

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Investigator's<br>Interpretation | Investigator's<br>Comment | Which AE the<br>Abnormality is<br>related to? | Which MH the<br>Abnormality is<br>related to? |
|---|---|---|---|---|---|---|---|
| S012/011 | Screening | 1st | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S012/011<br>S012/011 | Screening | 2nd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S012/011<br>S012/011 | Screening | 3rd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S012/011 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S012/011 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S012/011 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Normal | | | |
| S012/011 | End of study | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S012/011 | End of study | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S012/011 | End of study | 3rd | ddMMMyyyy hh:mm | Normal | | | |

Note: Subjects are listed according to the cohort they belong to

NCS: Not Clinically Significant Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.3 - Investigator's interpretation of ECG

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Investigator's<br>Interpretation | Investigator's<br>Comment | Which AE the<br>Abnormality is<br>related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|---|
| S024/021 | Screening | 1st | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S024/021 | Screening | 2nd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S024/021 | Screening | 3rd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S024/021 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S024/021 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S024/021 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Normal | | | |
| S024/021 | End of study | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S024/021 | End of study | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S024/021 | End of study | 3rd | ddMMMyyyy hh:mm | Normal | | | |

Note: Subjects are listed according to the cohort they belong to

NCS: Not Clinically Significant Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.3 - Investigator's interpretation of ECG

### Cohort 3: 5 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Investigator's<br>Interpretation | Investigator's<br>Comment | Which AE the<br>Abnormality is<br>related to? | Which MH the<br>Abnormality is<br>related to? |
|---|---|---|---|---|---|---|---|
| S036/031 | Screening | 1st | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| | • | | • • • • | , | | <del></del> | |
| S036/031 | Screening | 2nd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S036/031 | Screening | 3rd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S036/031 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S036/031 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S036/031 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Normal | | | |
| | | | | | <b></b> | | |
| S036/031 | End of study | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S036/031 | End of study | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S036/031 | End of study | 3rd | ddMMMyyyy hh:mm | Normal | | | |

Note: Subjects are listed according to the cohort they belong to

NCS: Not Clinically Significant Program: Listings\k363-eg-lst.sas



### Listing 16.2.9.3 - Investigator's interpretation of ECG

### Cohort 4: 2 min (T)

| Subject<br>ID | Time<br>Point | Replicate | Assessment<br>Date/Time | Investigator's<br>Interpretation | Investigator's<br>Comment | Which AE the<br>Abnormality is<br>related to? | Which MH the Abnormality is related to? |
|---|---|---|---|---|---|---|---|
| S048/041 | Screening | 1st | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S048/041 | Screening | 2nd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S048/041 | Screening | 3rd | ddMMMyyyy hh:mm | Abnormal, NCS | Irregularity in the heart rhythm | | |
| S048/041 | Visit 3 - Pre dose | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S048/041 | Visit 3 - Pre dose | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S048/041 | Visit 3 - Pre dose | 3rd | ddMMMyyyy hh:mm | Normal | | | |
| S048/041 | End of study | 1st | ddMMMyyyy hh:mm | Normal | | | |
| S048/041 | End of study | 2nd | ddMMMyyyy hh:mm | Normal | | | |
| S048/041 | End of study | 3rd | ddMMMyyyy hh:mm | Normal | | | |

Note: Subjects are listed according to the cohort they belong to

NCS: Not Clinically Significant Program: Listings\k363-eg-lst.sas



### Listing 16.2.10.1 - Medical and surgical history

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S001/001 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Date of Diagnosis: | JUL2019 |
| | | | Ongoing: | N |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Date of Surgery: | NOV1980 |
| | | ••• | ••• | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-mh-lst.sas



### Listing 16.2.10.1 - Medical and surgical history

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S012/011 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Date of Diagnosis: | JUL2019 |
| | | | Ongoing: | N |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Date of Surgery: | NOV1980 |
| | ••• | ••• | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-mh-lst.sas



### Listing 16.2.10.1 - Medical and surgical history

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S024/021 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Date of Diagnosis: | JUL2019 |
| | | | Ongoing: | N |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Date of Surgery: | NOV1980 |
| | | ••• | | ··· |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-mh-lst.sas



### Listing 16.2.10.1 - Medical and surgical history

### Cohort 3: 5 min (T)

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S036/031 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Date of Diagnosis: | JUL2019 |
| | | | Ongoing: | N |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Date of Surgery: | NOV1980 |
| | | | ••• | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-mh-lst.sas



### Listing 16.2.10.1 - Medical and surgical history

Cohort 4: 2 min (T)

| Subject<br>ID | Category | Disease/Surgery<br>ID | | |
|---|---|---|---|---|
| S048/041 | Medical History | M1 | Verbatim: | Left shoulder luxation |
| | | | Preferred Term 1: | Joint dislocation |
| | | | System Organ Class 1: | Injury, poisoning and procedural complications |
| | | | Date of Diagnosis: | JUL2019 |
| | | | Ongoing: | N |
| | Surgery | S1 | Verbatim: | Right knee meniscectomy |
| | | | Preferred Term 1: | Meniscus removal |
| | | | System Organ Class 1: | Surgical and medical procedures |
| | | | Date of Surgery: | NOV1980 |
| | | ••• | | ··· |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-mh-lst.sas



### Listing 16.2.10.2 - Physical examination

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S001/001 | Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | | ••• | | ••• |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Which AE (number) the Abnormality is related to? | 1 |
| | | | Which MH (number) the Abnormality is related to? | |
| | | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-pe-lst.sas



### Listing 16.2.10.2 - Physical examination

**Cohort 1: 30 min (T)** 

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S012/011 | Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Which AE (number) the Abnormality is related to? | 1 |
| | | | Which MH (number) the Abnormality is related to? | |
| | | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-pe-lst.sas



### Listing 16.2.10.2 - Physical examination

**Cohort 2: 15 min (T)** 

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S024/021 | Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | | | | ••• |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Which AE (number) the Abnormality is related to? | 1 |
| | | | Which MH (number) the Abnormality is related to? | |
| ••• | ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-pe-lst.sas



### Listing 16.2.10.2 - Physical examination

### Cohort 3: 5 min (T)

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S036/031 | Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Which AE (number) the Abnormality is related to? | 1 |
| | | | Which MH (number) the Abnormality is related to? | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-pe-lst.sas



### Listing 16.2.10.2 - Physical examination

# Cohort 4: 2 min (T)

| Subject<br>ID | Time Point | Physical<br>Examination<br>Date | | |
|---|---|---|---|---|
| S048/041 | Day -1 | ddMMMyyyy | Investigator's Interpretation | Normal |
| | ••• | | | |
| | End of Study | ddMMMyyyy | Investigator's Interpretation: | Abnormal, Clinically Significant |
| | | | Which AE (number) the Abnormality is related to? | 1 |
| | | | Which MH (number) the Abnormality is related to? | |
| | ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Note 1: MedDRA version 27.0 Program: Listings\k363-pe-lst.sas



### Listing 16.2.10.3 - Prior and concomitant medications

#### **Cohort 1: 30 min (Rα)**

| Subject<br>ID | Category | Medication<br>ID | | |
|---|---|---|---|---|
| S001/001 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class <sup>1, 2</sup> : | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose per Administration: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |

Note: Subjects are listed according to the cohort they belong to

Note 1: WHO Drug Dictionary Enhanced March 1, 2024

Note 2: Anatomical Therapeutic Chemical classification, 4th level term

Program: Listings\k363-cm-lst.sas



### Listing 16.2.10.3 - Prior and concomitant medications

### **Cohort 1: 30 min (T)**

| Subject<br>ID | Category | Medication<br>ID | | |
|---|---|---|---|---|
| S012/011 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class <sup>1, 2</sup> : | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose per Administration: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class 1, 2: | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |

Note: Subjects are listed according to the cohort they belong to

Note 1: WHO Drug Dictionary Enhanced March 1, 2024

Note 2: Anatomical Therapeutic Chemical classification, 4th level term  $\,$ 

Program: Listings\k363-cm-lst.sas



### Listing 16.2.10.3 - Prior and concomitant medications

### **Cohort 2: 15 min (T)**

| Subject<br>ID | Category | Medication<br>ID | | |
|---|---|---|---|---|
| S024/021 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class <sup>1, 2</sup> : | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose per Administration: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class 1, 2: | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |

Note: Subjects are listed according to the cohort they belong to

Note 1: WHO Drug Dictionary Enhanced March 1, 2024

Note 2: Anatomical Therapeutic Chemical classification, 4th level term  $\,$ 

Program: Listings\k363-cm-lst.sas


## Listing 16.2.10.3 - Prior and concomitant medications

## Cohort 3: 5 min (T)

| Subject<br>ID | Category | Medication ID | | |
|---|---|---|---|---|
| S036/031 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class <sup>1, 2</sup> : | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose per Administration: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |

Note: Subjects are listed according to the cohort they belong to

Note 1: WHO Drug Dictionary Enhanced March 1, 2024

Note 2: Anatomical Therapeutic Chemical classification, 4th level term  $\,$ 

Program: Listings\k363-cm-lst.sas



## Listing 16.2.10.3 - Prior and concomitant medications

## Cohort 4: 2 min (T)

| Subject<br>ID | Category | Medication ID | | |
|---|---|---|---|---|
| S048/041 | Prior | 1 | Verbatim: | Alerid |
| | | | Standardised Medication Name 1: | Alerid |
| | | | Active Ingredients 1: | Cetirizine hydrochloride |
| | | | Medication Class <sup>1, 2</sup> : | Piperazine derivatives (R06AE) |
| | | | Indication: | Pollinosis |
| | | | Dose per Administration: | 10 mg |
| | | | Start - End Date/Time: | 2013 - Ongoing |
| | | | Frequency - Route: | 1 time per day - Oral |
| | Concomitant | 2 | Verbatim: | Paracen |
| | | | Standardised Medication Name 1: | Paracen |
| | | | Active Ingredients 1: | Paracetamol |
| | | | Medication Class <sup>1, 2</sup> : | Anilides (N02BE) |
| | | | Indication: | Headache |
| | | | Dose: | 500 mg |
| | | | Start - End Date/Time: | 15JUN2019 19:08 - 15JUN2019 19:08 |
| | | | Frequency - Route: | Once - Oral |

Note: Subjects are listed according to the cohort they belong to

Note 1: WHO Drug Dictionary Enhanced March 1, 2024

Note 2: Anatomical Therapeutic Chemical classification, 4th level term  $\,$ 

Program: Listings\k363-cm-lst.sas



#### Listing 16.2.10.4 - Substance use

#### **Cohort 1: 30 min (Rα)**

| Subject ID | Category | Consumption level | Consumption per Day | <b>End of consumption Date</b> |
|---|---|---|---|---|
| S001/001 | Tobacco | Non smoker | | |
| | Alcohol | Occasionally | | |
| | Caffeine | No consumption | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-su-lst.sas



#### Listing 16.2.10.4 - Substance use

**Cohort 1: 30 min (T)** 

| Subject ID | Category | Consumption level | <b>Consumption per Day</b> | <b>End of consumption Date</b> |
|---|---|---|---|---|
| S012/011 | Tobacco | Ex smoker | | JUL2018 |
| | Alcohol | Regularly | 4 drinks per day | |
| | Caffeine | Consumption | 3 cups coffee/tea per day | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-su-lst.sas



#### Listing 16.2.10.4 - Substance use

**Cohort 2: 15 min (T)** 

| Subject ID | Category | <b>Consumption level</b> | Consumption per Day | <b>End of consumption Date</b> |
|---|---|---|---|---|
| S024/021 | Tobacco | Smoker | 10 cigarettes per day | |
| | Alcohol | Occasionally | | |
| | Caffeine | Consumption | 5 cups coffee/tea per day | |
| ··· | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-su-lst.sas



#### Listing 16.2.10.4 - Substance use

# Cohort 3: 5 min (T)

| Subject ID | Category | <b>Consumption level</b> | <b>Consumption per Day</b> | <b>End of consumption Date</b> |
|---|---|---|---|---|
| S036/031 | Tobacco | Smoker | 5 cigarettes per day | |
| | Alcohol | No | | |
| | Caffeine | No consumption | <del></del> | <del></del> |
| ••• | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-su-lst.sas



#### Listing 16.2.10.4 - Substance use

# Cohort 4: 2 min (T)

| Subject ID | Category | Consumption level | Consumption per Day | <b>End of consumption Date</b> |
|---|---|---|---|---|
| S048/041 | Tobacco | Non smoker | | |
| | Alcohol | No | | |
| | Caffeine | Consumption | 5 cups coffee/tea per day | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-su-lst.sas



## Listing 16.2.10.5 - Subjects study visits

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | Screening Visit 1 Day -14/-2 | Visit 2<br>Day -1<br>Date (Day) | Visit 3<br>Day 1<br>Start Date (Day) | Visit 3<br>Day 2<br>End Date (Day) | Final Visit<br>Visit 4<br>Date (Day) | Early Termination<br>Visit<br>Date (Day) |
|---|---|---|---|---|---|---|
| S001/001 | Date (Day) ddMMMyyyy (-j) | ddMMMyyyy (-1)<br> | ddMMMyyyy (1) | ddMMMyyyy (1) | ddMMMyyyy (6) | ddMMMyyyy (x) |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-sv-lst.sas



## Listing 16.2.10.5 - Subjects study visits

**Cohort 1: 30 min (T)** 

| Subject | Screening | Visit 2 | Visit 3 | Visit 3 | Final Visit | <b>Early Termination</b> |
|---|---|---|---|---|---|---|
| ID | Visit 1 | <b>Day -1</b> | Day 1 | Day 2 | Visit 4 | Visit |
| | <b>Day -14/-2</b> | Date (Day) | Start Date (Day) | End Date (Day) | Date (Day) | Date (Day) |
| | Date (Day) | | | | | |
| S012/011 | ddMMMyyyy (-j) | ddMMMyyyy (-1) | ddMMMyyyy (1) | ddMMMyyyy (1) | ddMMMyyyy (6) | ddMMMyyyy (x) |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-sv-lst.sas



## Listing 16.2.10.5 - Subjects study visits

**Cohort 2: 15 min (T)** 

| Subject | Screening | Visit 2 | Visit 3 | Visit 3 | Final Visit | Early Termination |
|---|---|---|---|---|---|---|
| ID | Visit 1 | <b>Day -1</b> | Day 1 | Day 2 | Visit 4 | Visit |
| | Day -14/-2 | Date (Day) | Start Date (Day) | End Date (Day) | Date (Day) | Date (Day) |
| | Date (Day) | | | | | |
| S024/021 | ddMMMyyyy (-j) | ddMMMyyyy (-1) | ddMMMyyyy (1) | ddMMMyyyy (1) | ddMMMyyyy (6) | ddMMMyyyy (x) |
| | ••• | ••• | | ••• | ••• | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-sv-lst.sas



## Listing 16.2.10.5 - Subjects study visits

Cohort 3: 5 min (T)

| Subject | Screening | Visit 2 | Visit 3 | Visit 3 | Final Visit | <b>Early Termination</b> |
|---|---|---|---|---|---|---|
| ID | Visit 1 | <b>Day -1</b> | Day 1 | Day 2 | Visit 4 | Visit |
| | <b>Day -14/-2</b> | Date (Day) | Start Date (Day) | End Date (Day) | Date (Day) | Date (Day) |
| | Date (Day) | | | | | |
| S036/031 | ddMMMyyyy (-j) | ddMMMyyyy (-1) | ddMMMyyyy (1) | ddMMMyyyy (1) | ddMMMyyyy (6) | ddMMMyyyy (x) |
| ••• | ••• | ••• | | | | ••• |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-sv-lst.sas



## Listing 16.2.10.5 - Subjects study visits

Cohort 4: 2 min (T)

| Subject | Screening | Visit 2 | Visit 3 | Visit 3 | Final Visit | Early Termination |
|---|---|---|---|---|---|---|
| ID | Visit 1 | <b>Day -1</b> | Day 1 | Day 2 | Visit 4 | Visit |
| | <b>Day -14/-2</b> | Date (Day) | Start Date (Day) | End Date (Day) | Date (Day) | Date (Day) |
| | Date (Day) | | | | | |
| S048/041 | ddMMMyyyy (-j) | ddMMMyyyy (-1) | ddMMMyyyy (1) | ddMMMyyyy (1) | ddMMMyyyy (6) | ddMMMyyyy (x) |
| | ••• | | | ••• | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-sv-lst.sas



## Listing 16.2.10.6 - Fertility status and contraception

#### **Cohort 1: 30 min (Rα)**

| Subject ID | Chilbearing Potential? | Reason for not childbearing potential? | Reliable Contraceptive Method Used? |
|---|---|---|---|
| S002/001 | Yes | <del></del> | Yes |
| ••• | <b></b> | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Only female subjects are listed Program: Listings\k363-rp-lst.sas



## Listing 16.2.10.6 - Fertility status and contraception

**Cohort 1: 30 min (T)** 

| Subject ID | Chilbearing Potential? | Reason for not childbearing potential? | Reliable Contraceptive Method Used? |
|---|---|---|---|
| S013/012 | Yes | <del></del> | Yes |
| | ··· | | |

Note: Subjects are listed according to the cohort they belong to

Only female subjects are listed

Program: Listings\k363-rp-lst.sas



## Listing 16.2.10.6 - Fertility status and contraception

**Cohort 2: 15 min (T)** 

| Subject ID | Chilbearing Potential? | Reason for not childbearing potential? | Reliable Contraceptive Method Used? |
|---|---|---|---|
| S025/022 | No | Surgical Sterilisation | |

Note: Subjects are listed according to the cohort they belong to

Only female subjects are listed

Program: Listings\k363-rp-lst.sas



## Listing 16.2.10.6 - Fertility status and contraception

## Cohort 3: 5 min (T)

| Subject ID | Chilbearing Potential? | Reason for not childbearing potential? | Reliable Contraceptive Method Used? |
|---|---|---|---|
| S036/031 | Yes | <del></del> | Yes |
| ••• | | | |

Note: Subjects are listed according to the cohort they belong to

Only female subjects are listed

Program: Listings\k363-rp-lst.sas



## Listing 16.2.10.6 - Fertility status and contraception

Cohort 4: 2 min (T)

| Subject ID | Chilbearing Potential? | Reason for not childbearing potential? | Reliable Contraceptive Method Used? |
|---|---|---|---|
| S049/042 | No | 12 months of spontaneous amenorrhea | |
| | | <b></b> | |

Note: Subjects are listed according to the cohort they belong to

Only female subjects are listed

Program: Listings\k363-rp-lst.sas



#### Listing 16.2.10.7 - Reproductive status and contraception

**Cohort 1: 30 min (Rα)** 

| Subject ID | Is he Sterile? | Approved Contraceptive Method Used? |
|------------|----------------|-------------------------------------|
| S002/001 | No | Yes |
| ••• | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Only male subjects are listed Program: Listings\k363-rp-lst.sas



#### Listing 16.2.10.7 - Reproductive status and contraception

**Cohort 1: 30 min (T)** 

| Subject ID | Is he Sterile? | Approved Contraceptive Method Used? |
|------------|----------------|-------------------------------------|
| S012/011 | Ye | <del></del> |

Note: Subjects are listed according to the cohort they belong to

Only male subjects are listed Program: Listings\k363-rp-lst.sas



#### Listing 16.2.10.7 - Reproductive status and contraception

**Cohort 2: 15 min (T)** 

| Subject ID | Is he Sterile? | Approved Contraceptive Method Used? |
|------------|----------------|-------------------------------------|
| S024/021 | No | Yes |
| ••• | | |

Note: Subjects are listed according to the cohort they belong to

Only male subjects are listed Program: Listings\k363-rp-lst.sas



#### Listing 16.2.10.7 - Reproductive status and contraception

Cohort 3: 5 min (T)

| Subject ID | Is he Sterile? | Approved Contraceptive Method Used? |
|------------|----------------|-------------------------------------|
| S036/031 | Ye | <del></del> |
| ••• | | <b></b> |

Note: Subjects are listed according to the cohort they belong to

Only male subjects are listed Program: Listings\k363-rp-lst.sas



#### Listing 16.2.10.7 - Reproductive status and contraception

Cohort 4: 2 min (T)

| Subject ID | Is he Sterile? | Approved Contraceptive Method Used? |
|------------|----------------|-------------------------------------|
| S049/042 | No | Yes |

Note: Subjects are listed according to the cohort they belong to

Only male subjects are listed Program: Listings\k363-rp-lst.sas



**Listing 16.2.10.8 - Meals** 

**Cohort 1: 30 min (Rα)** 

| Subject<br>ID | IMP Administration<br>Date/Time | Meal<br>Number | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/Time |
|---|---|---|---|---|---|---|
| S001/001 | ddMMMyyyy hh:mm | 1 | Dinner | Visit 2 - Day -1 | Y | ddMMMyyyy hh:mm |
| S001/001 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 - 5 hours post-dose | Y | ddMMMyyyy hh:mm |
| S001/001 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 - 12 hours post-dose | Y | ddMMMyyyy hh:mm |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ml-lst.sas



**Listing 16.2.10.8 - Meals** 

**Cohort 1: 30 min (T)** 

| Subject<br>ID | IMP Administration<br>Date/Time | Meal<br>Number | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/Time |
|---|---|---|---|---|---|---|
| S012/011 | ddMMMyyyy hh:mm | 1 | Dinner | Visit 2 - Day -1 | Y | ddMMMyyyy hh:mm |
| S012/011 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 - 5 hours post-dose | Y | ddMMMyyyy hh:mm |
| S012/011 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 - 12 hours post-dose | Y | ddMMMyyyy hh:mm |
| ••• | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ml-lst.sas



**Listing 16.2.10.8 - Meals** 

**Cohort 2: 15 min (T)** 

| Subject<br>ID | IMP Administration<br>Date/Time | Meal<br>Number | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/Time |
|---|---|---|---|---|---|---|
| S024/021 | ddMMMyyyy hh:mm | 1 | Dinner | Visit 2 - Day -1 | Y | ddMMMyyyy hh:mm |
| S024/021 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 - 5 hours post-dose | Y | ddMMMyyyy hh:mm |
| S024/021 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 - 12 hours post-dose | Y | ddMMMyyyy hh:mm |
| ••• | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ml-lst.sas



## **Listing 16.2.10.8 - Meals**

Cohort 3: 5 min (T)

| Subject<br>ID | IMP Administration Date/Time | Meal<br>Number | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/Time |
|---|---|---|---|---|---|---|
| S036/031 | ddMMMyyyy hh:mm | 1 | Dinner | Visit 2 - Day -1 | Y | ddMMMyyyy hh:mm |
| S036/031 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 - 5 hours post-dose | Y | ddMMMyyyy hh:mm |
| S036/031 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 - 12 hours post-dose | Y | ddMMMyyyy hh:mm |
| ••• | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ml-lst.sas



## **Listing 16.2.10.8 - Meals**

Cohort 4: 2 min (T)

| Subject<br>ID | IMP Administration Date/Time | Meal<br>Number | Standardised<br>Meal | Time Point | Meal<br>Served? | Meal Start<br>Date/Time |
|---|---|---|---|---|---|---|
| S048/041 | ddMMMyyyy hh:mm | 1 | Dinner | Visit 2 - Day -1 | Y | ddMMMyyyy hh:mm |
| S048/041 | ddMMMyyyy hh:mm | 2 | Lunch | Day 1 - 5 hours post-dose | Y | ddMMMyyyy hh:mm |
| S048/041 | ddMMMyyyy hh:mm | 3 | Dinner | Day 1 - 12 hours post-dose | Y | ddMMMyyyy hh:mm |
| ••• | | | | | | |

Note: Subjects are listed according to the cohort they belong to

Program: Listings\k363-ml-lst.sas